CLINICAL TRIAL: NCT02780167
Title: A PHASE 2B RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, PARALLEL, MULTICENTER, DOSE-RANGING, STUDY TO EVALUATE THE EFFICACY AND SAFETY PROFILE OF PF-04965842 IN SUBJECTS WITH MODERATE TO SEVERE ATOPIC DERMATITIS
Brief Title: Study To Evaluate Pf-04965842 In Subjects With Moderate To Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B7451006; 2015-005513-72 (EudraCT Number)
Record Dates: First submitted 2016-04-11; First posted 2016-05-23 (Estimated); Results first posted 2018-05-16 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Atopic Dermatitis
Keywords: Phase 2; randomized; double-blind; placebo; atopic dermatitis; safety; efficacy; JAK; janus kinase; moderate; severe
MeSH Terms: conditions — Dermatitis, Atopic; Lymphoma, Follicular | interventions — abrocitinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1 (Experimental): 10 mg of PF-04965842 QD
  Interventions: Drug: PF-04965842
- Cohort 2 (Experimental): 30 mg of PF-04965842 QD
  Interventions: Drug: PF-04965842
- Cohort 3 (Experimental): 100 mg of PF-04965842 QD
  Interventions: Drug: PF-04965842
- Cohort 4 (Experimental): 200 mg of PF-04965842 QD
  Interventions: Drug: PF-04965842
- Cohort 5 (Placebo Comparator): placebo QD
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-04965842 — 10 mg of PF-04965842 QD for 12 weeks
  Arms: Cohort 1
Drug: PF-04965842 — 30 mg of PF-04965842 QD for 12 weeks
  Arms: Cohort 2
Drug: PF-04965842 — 100 mg of PF-04965842 QD for 12 weeks
  Arms: Cohort 3
Drug: PF-04965842 — 200 mg of PF-04965842 QD for 12 weeks
  Arms: Cohort 4
Drug: Placebo — Placebo QD for 12 weeks
  Arms: Cohort 5

SUMMARY:
Study B7451006 is a Phase 2b POC study which is planned to assess four PF 04965842 once daily (QD) doses (10, 30, 100, 200 mg) relative to placebo over 12 weeks to characterize the efficacy and safety of PF 04965842 in subjects with moderate to severe AD. The objectives of the study are to demonstrate the efficacy of PF 04965842 by showing improvement in disease severity in patients with moderate to severe AD as measured by the Investigator's Global Assessment (IGA) and Eczema Area and Severity Index (EASI) scores, and safety to support further clinical development of PF 04965842.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between 18 75 years of age, inclusive, at time of informed consent.
* Must have the following atopic dermatitis criteria:

  1. Have a clinical diagnosis of chronic atopic dermatitis (also known as atopic eczema) for at least 1 year prior to Day 1 and has confirmed atopic dermatitis (Hanifin and Rajka criteria of AD refer to Appendix 2) at the Screening visit.
  2. Have inadequate response to treatment with topical medications given for at least 4 weeks, or for whom topical treatments are otherwise medically inadvisable (eg, because of important side effects or safety risks) within 12 months of the first dose of study drug.
  3. Moderate to severe AD (affected BSA >=10 %, IGA >=3, and EASI >=12 at the screening and baseline visits).

Exclusion Criteria:

* History of human immunodeficiency virus (HIV) or positive HIV serology at screening,
* Infected with hepatitis B or hepatitis C viruses.
* Have evidence of active or latent or inadequately treated infection with Mycobacterium tuberculosis (TB)
* Have received any of the following treatment regiments specified in the timeframes outlined below:

Within 6 months of first dose of study drug: Any cell depleting agents Within 12 weeks of first dose of study drug: Any studies with JAK inhibitors; Other biologics Within 8 weeks of first dose of study drug: Participation in other studies involving investigational drug(s) Within 6 weeks of first dose of study drug: Have been vaccinated with live or attenuated live vaccine.

Within 4 weeks of first dose of study drug: Use of oral immune suppressants; Phototherapy (NB UVB) or broad band phototherapy; Regular use (more than 2 visits per week) of a tanning booth/parlor.

Within 1 week of first dose of study drug: Topical treatments that could affect atopic dermatitis; Herbal medications with unknown properties or known beneficial effects for AD.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (64):
- United States (37):
  - Clinical Research Center of Alabama, Birmingham, Alabama
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - Huntington Medical Foundation, Pasadena, California
  - Peninsula Research Associates, Inc., Rolling Hills Estates, California
  - Emil A. Tanghetti MD dba Center for Dermatology and Laser Surgery, Sacramento, California
  - TCR Medical Corporation, San Diego, California
  - Clinical Science Institute, Santa Monica, California
  - University of Connecticut Health Center (UConn Health), Farmington, Connecticut
  - Olympian Clinical Research, Clearwater, Florida
  - North Florida Dermatology Associates, PA, Jacksonville, Florida
  - Park Avenue Dermatology Administration Annex, Orange Park, Florida
  - Park Avenue Dermatology, Orange Park, Florida
  - Leavitt Medical Associates of Florida d/b/a Ameriderm Research, Ormond Beach, Florida
  - Forward Clinical Trials, Inc., Tampa, Florida
  - MedaPhase, Inc., Newnan, Georgia
  - Dundee Dermatology, West Dundee, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Dawes Fretzin Dermatology Group, LLC, Indianapolis, Indiana
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - DS Research, Louisville, Kentucky
  - Shondra L Smith, MD Dermatology & Advanced Aesthetics, Lake Charles, Louisiana
  - Somerset Skin Centre, Troy, Michigan
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - Clinical Research Consortium, Las Vegas, Nevada
  - Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey
  - The Dermatology Group, P.C, Verona, New Jersey
  - Forest Hills Dermatology Group, Forest Hills, New York
  - Sadick Research Group, New York, New York
  - Vital Prospects Clinical Research Institute, P.C, Tulsa, Oklahoma
  - DermDox Centers for Dermatology, Hazleton, Pennsylvania
  - UPMC Department of Dermatology, Pittsburgh, Pennsylvania
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Health Concepts, Rapid City, South Dakota
  - Bellaire Dermatology Associates, Bellaire, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Virginia Clinical Research,Inc, Norfolk, Virginia
  - West End Dermatology Associates, Richmond, Virginia
- Australia (8):
  - Woden Dermatology, Phillip, Australian Capital Territory
  - Australian Clinical Research Network, Sydney, New South Wales
  - The Skin Centre, Benowa, Queensland
  - Veracity Clinical Research, Woolloongabba, Queensland
  - Sinclair Dermatology, East Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Fremantle Dermatology, Fremantle, Western Australia
  - North Eastern Health Specialists, Hectorville, South Australia
- Canada (11):
  - University of British Columbia, Vancouver, British Columbia
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - Lynderm Research Inc., Markham, Ontario
  - Research by ICLS, Oakville, Ontario
  - Skin Centre for Dermatology, Peterborough, Ontario
  - The Centre for Dermatology, Richmond Hill, Ontario
  - K. Papp Clinical Research, Waterloo, Ontario
  - Windsor Clinical Research Inc, Windsor, Ontario
  - Innovaderm Research Inc., Montreal, Quebec
  - Centre de Recherche Dermatologique du Quebec metropolitain (CRDQ), Québec, Quebec
  - Diex Research Sherbrooke Inc., Sherbrooke, Quebec
- Germany (4):
  - ISA GmbH, Berlin
  - Universitaetsklinikum Schleswig-Holstein, Lübeck
  - Universitaetsklinikum Muenster, Münster
  - Universitaetsklinikum Tuebingen, Tübingen
- Hungary (4):
  - Bacs Kiskun Megyei Korhaz, Bor es Nemibeteggondozo, Kecskemét
  - CRU Hungary Ltd., MISEK-CRU, Miskolc
  - Szegedi Tudomanyegyetem SzentGyorgyi Albert Klinikai Kozpont Borgyogyaszati es Allergologiai Klinika, Szeged
  - Allergo-Derm Bakos Kft., Szolnok

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Silverberg JI, Thyssen JP, Lazariciu I, Myers DE, Guler E, Chovatiya R. Abrocitinib may improve itch and quality of life in patients with itch-dominant atopic dermatitis. Skin Health Dis. 2024 May 5;4(4):e382. doi: 10.1002/ski2.382. eCollection 2024 Aug. PMID 39104653
- [Derived] Armstrong AW, Alexis AF, Blauvelt A, Silverberg JI, Feeney C, Levenberg M, Chan G, Zhang F, Fostvedt L. Predicting Abrocitinib Efficacy at Week 12 Based on Clinical Response at Week 4: A Post Hoc Analysis of Four Randomized Studies in Moderate-to-Severe Atopic Dermatitis. Dermatol Ther (Heidelb). 2024 Jul;14(7):1849-1861. doi: 10.1007/s13555-024-01183-3. Epub 2024 Jun 19. PMID 38896380
- [Derived] Schmid-Grendelmeier P, Gooderham MJ, Hartmann K, Konstantinou GN, Fellmann M, Koulias C, Clibborn C, Biswas P, Brunner PM. Efficacy and safety of abrocitinib in patients with moderate-to-severe atopic dermatitis and comorbid allergies. Allergy. 2024 Jan;79(1):174-183. doi: 10.1111/all.15952. Epub 2023 Nov 21. PMID 37988255
- [Derived] Alexis AF, Silverberg JI, Rice ZP, Armstrong AW, Desai SR, Fonacier L, Kabashima K, Biswas P, Cella RR, Chan GL, Levenberg M. Abrocitinib efficacy and safety in moderate-to-severe atopic dermatitis by race, ethnicity, and Fitzpatrick skin type. Ann Allergy Asthma Immunol. 2024 Mar;132(3):383-389.e3. doi: 10.1016/j.anai.2023.11.002. Epub 2023 Nov 10. PMID 37949351
- [Derived] Gooderham MJ, Girolomoni G, Moore JO, Silverberg JI, Bissonnette R, Forman S, Peeva E, Biswas P, Valdez H, Chan G. Durability of Response to Abrocitinib in Patients with Moderate-to-Severe Atopic Dermatitis After Treatment Discontinuation in a Phase 2b Trial. Dermatol Ther (Heidelb). 2022 Sep;12(9):2077-2085. doi: 10.1007/s13555-022-00764-4. Epub 2022 Aug 7. PMID 35933552
- [Derived] Blauvelt A, Boguniewicz M, Brunner PM, Luna PC, Biswas P, DiBonaventura M, Farooqui SA, Rojo R, Cameron MC. Abrocitinib monotherapy in Investigator's Global Assessment nonresponders: improvement in signs and symptoms of atopic dermatitis and quality of life. J Dermatolog Treat. 2022 Aug;33(5):2605-2613. doi: 10.1080/09546634.2022.2059053. Epub 2022 Jul 6. PMID 35763326
- [Derived] Stander S, Bhatia N, Gooderham MJ, Silverberg JI, Thyssen JP, Biswas P, DiBonaventura M, Romero W, Farooqui SA. High threshold efficacy responses in moderate-to-severe atopic dermatitis are associated with additional quality of life benefits: pooled analyses of abrocitinib monotherapy studies in adults and adolescents. J Eur Acad Dermatol Venereol. 2022 Aug;36(8):1308-1317. doi: 10.1111/jdv.18170. Epub 2022 May 6. PMID 35462428
- [Derived] Wojciechowski J, Malhotra BK, Wang X, Fostvedt L, Valdez H, Nicholas T. Population pharmacokinetic-pharmacodynamic modelling of platelet time-courses following administration of abrocitinib. Br J Clin Pharmacol. 2022 Aug;88(8):3856-3871. doi: 10.1111/bcp.15334. Epub 2022 Apr 11. PMID 35342978
- [Derived] Wojciechowski J, Malhotra BK, Wang X, Fostvedt L, Valdez H, Nicholas T. Population Pharmacokinetics of Abrocitinib in Healthy Individuals and Patients with Psoriasis or Atopic Dermatitis. Clin Pharmacokinet. 2022 May;61(5):709-723. doi: 10.1007/s40262-021-01104-z. Epub 2022 Jan 21. PMID 35061234
- [Derived] Simpson EL, Silverberg JI, Nosbaum A, Winthrop KL, Guttman-Yassky E, Hoffmeister KM, Egeberg A, Valdez H, Zhang M, Farooqui SA, Romero W, Thorpe AJ, Rojo R, Johnson S. Integrated Safety Analysis of Abrocitinib for the Treatment of Moderate-to-Severe Atopic Dermatitis From the Phase II and Phase III Clinical Trial Program. Am J Clin Dermatol. 2021 Sep;22(5):693-707. doi: 10.1007/s40257-021-00618-3. Epub 2021 Aug 18. PMID 34406619
- [Derived] Silverberg JI, Thyssen JP, Simpson EL, Yosipovitch G, Stander S, Valdez H, Rojo R, Biswas P, Myers DE, Feeney C, DiBonaventura M. Impact of Oral Abrocitinib Monotherapy on Patient-Reported Symptoms and Quality of Life in Adolescents and Adults with Moderate-to-Severe Atopic Dermatitis: A Pooled Analysis of Patient-Reported Outcomes. Am J Clin Dermatol. 2021 Jul;22(4):541-554. doi: 10.1007/s40257-021-00604-9. Epub 2021 May 5. PMID 33954933
- [Derived] Simpson EL, Wollenberg A, Bissonnette R, Silverberg JI, Papacharalambous J, Zhu L, Zhang W, Beebe JS, Vincent M, Peeva E, Bushmakin AG, Cappelleri JC, Chen L, Sikirica V, Xenakis J. Patient-Reported Symptoms and Disease Impacts in Adults With Moderate-to-Severe Atopic Dermatitis: Results From a Phase 2b Study With Abrocitinib. Dermatitis. 2021 Oct 1;32(1S):S53-S61. doi: 10.1097/DER.0000000000000725. PMID 33795561
- [Derived] Gooderham MJ, Forman SB, Bissonnette R, Beebe JS, Zhang W, Banfield C, Zhu L, Papacharalambous J, Vincent MS, Peeva E. Efficacy and Safety of Oral Janus Kinase 1 Inhibitor Abrocitinib for Patients With Atopic Dermatitis: A Phase 2 Randomized Clinical Trial. JAMA Dermatol. 2019 Dec 1;155(12):1371-1379. doi: 10.1001/jamadermatol.2019.2855. PMID 31577341
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7451006&StudyName=A+Phase+2b+Randomized%2C+Double%E2%80%91blind%2C+Placebo-controlled%2C+Parallel%2C+Multicenter%2C+Dose-ranging%2C+Study+To+Evaluate+The+Efficacy+And+Safety+Profile+Of+Pf-04965842+In+Subjects+With+Moderate+To+Severe+Atopic+Dermatitis

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 269 participants were randomized. There were 2 participants who were randomized but did not receive any study treatment. All other participants were treated.
Groups:
- Placebo: Participants received matching placebo tablets for a 12-week double-blind treatment period.
- PF-04965842 10mg QD: Participants received PF-04965842 10 mg once daily for a 12-week double-blind treatment period.
- PF-04965842 30mg QD: Participants received PF-04965842 30 mg once daily for a 12-week double-blind treatment period.
- PF-04965842 100mg QD: Participants received PF-04965842 100 mg once daily for a 12-week double-blind treatment period.
- PF-04965842 200mg QD: Participants received PF-04965842 200 mg once daily for a 12-week double-blind treatment period.
Period: Overall Study
Arm/Group | Placebo | PF-04965842 10mg QD | PF-04965842 30mg QD | PF-04965842 100mg QD | PF-04965842 200mg QD
Started | 56 | 49 | 51 | 56 | 55
Completed | 28 | 27 | 27 | 37 | 38
Not Completed | 28 | 22 | 24 | 19 | 17
Not completed — Adverse Event | 9 | 8 | 8 | 12 | 8
Not completed — Lack of Efficacy | 6 | 5 | 6 | 1 | 0
Not completed — Lost to Follow-up | 2 | 0 | 1 | 0 | 0
Not completed — Does not meet entrance criteria | 0 | 0 | 1 | 0 | 0
Not completed — No longer meets eligibility criteria | 0 | 0 | 0 | 1 | 1
Not completed — Protocol Violation | 5 | 5 | 1 | 1 | 2
Not completed — Withdrawal by Subject | 6 | 4 | 4 | 3 | 4
Not completed — Other | 0 | 0 | 3 | 1 | 2

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) was defined as all randomized participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-04965842 10mg QD | PF-04965842 30mg QD | PF-04965842 100mg QD | PF-04965842 200mg QD | Total
Number analyzed (Participants) | 56 | 49 | 51 | 56 | 55 | 267
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (15.1) | 44.3 (15.9) | 37.6 (15.9) | 41.1 (15.6) | 38.7 (17.6) | 40.8 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 28 | 29 | 25 | 27 | 144
  Male | 21 | 21 | 22 | 31 | 28 | 123
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 40 | 38 | 39 | 40 | 37 | 194
  Black | 10 | 5 | 4 | 7 | 13 | 39
  Asian | 4 | 5 | 5 | 8 | 5 | 27
  Other | 2 | 1 | 3 | 1 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving the Investigator's Global Assessment (IGA) for Clear (0) or Almost Clear (1) and >=2 Points Improvement From Baseline at Week 12
Description: The IGA score quantifies the severity of participants' atopic dermatitis (AD). Scores range from 0 to 4 and correspond to a category (clear, almost clear, mild, moderate and severe, respectively).
Time Frame: Baseline and Week 12
Population: "Number of Participants Analyzed" represents the number of participants in the full analysis set (FAS) population. "Number Analyzed" at each visit represents the number of evaluable subjects for that visit.
Measure: Least Squares Mean (Standard Error); unit: percentage of participants
Arm/Group | Placebo | PF-04965842 10mg QD | PF-04965842 30mg QD | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 56 | 49 | 51 | 56 | 55
percentage of participants | 6.3 (2.55) | 8.2 (2.32) | 12.3 (2.88) | 27.8 (5.07) | 44.5 (6.92)
Statistical Analysis 1: Comparison: Placebo vs PF-04965842 10mg QD; Test type: Other; p = 0.1210, Emax model; Emax model with non-responder imputation (NRI); Estimate difference = 1.8, 95% CI 2-sided [-0.7 to 4.4], Standard Error of Mean 0.99 — Test group: PF-04965842 10 mg QD, Reference group: Placebo
Statistical Analysis 2: Comparison: Placebo vs PF-04965842 30mg QD; Test type: Other; p = 0.1065, Emax model; Emax model with non-responder imputation (NRI); Estimate difference = 6.0, 95% CI 2-sided [-1.8 to 13.8], Standard Error of Mean 3.05 — Test group: PF-04965842 30 mg QD, Reference group: Placebo
Statistical Analysis 3: Comparison: Placebo vs PF-04965842 100mg QD; Test type: Other; p = 0.0184, Emax model; Emax model with non-responder imputation (NRI); Estimate difference = 21.5, 95% CI 2-sided [5.5 to 37.6], Standard Error of Mean 6.25 — Test group: PF-04965842 100 mg QD, Reference group: Placebo
Statistical Analysis 4: Comparison: Placebo vs PF-04965842 200mg QD; Test type: Other; p = 0.0032, Emax model; Emax model with non-responder imputation (NRI); Mean Difference (Final Values) = 38.2, 95% CI 2-sided [19.7 to 56.6], Standard Error of Mean 7.18 — Test group: PF-04965842 200 mg QD, Reference group: Placebo

2. Secondary Outcome: Percent Change From Baseline in the Eczema Area and Severity Index (EASI) at Week 12
Description: The EASI quantifies the severity of participants' AD based on both severity of lesion clinical signs and the percent of body surface area (BSA) affected. EASI is a composite scoring by the AD clinical evaluator of the degree of erythema, induration/population, excoriation, and lichenification (each scored separately) for each of 4 regions, with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The EASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of AD.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | PF-04965842 10mg QD | PF-04965842 30mg QD | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 56 | 49 | 51 | 56 | 55
percent change | -35.22 (6.572) | -31.13 (7.090) | -40.73 (6.823) | -59.04 (6.212) | -82.57 (6.161)
Statistical Analysis 1: Comparison: Placebo vs PF-04965842 10mg QD; Test type: Other; p = 0.6731, Mixed Models Analysis; Mixed-effects model repeated measures (MMRM) with observed cases (OC); LS mean difference = 4.08, 90% CI 2-sided [-11.88 to 20.05], Standard Error of Mean 9.667 — Test group: PF-04965842 10 mg QD, Reference group: Placebo
Statistical Analysis 2: Comparison: Placebo vs PF-04965842 30mg QD; Test type: Other; p = 0.5610, Mixed Models Analysis; MMRM with OC; LS mean difference = -5.52, 90% CI 2-sided [-21.16 to 10.13], Standard Error of Mean 9.474 — Test group: PF-04965842 30 mg QD, Reference group: Placebo
Statistical Analysis 3: Comparison: Placebo vs PF-04965842 100mg QD; Test type: Other; p = 0.0091, Mixed Models Analysis; MMRM with OC; LS mean difference = -23.82, 90% CI 2-sided [-38.76 to -8.88], Standard Error of Mean 9.043 — Test group: PF-04965842 100 mg QD, Reference group: Placebo
Statistical Analysis 4: Comparison: Placebo vs PF-04965842 200mg QD; Test type: Other; p < 0.0001, Mixed Models Analysis; MMRM with OC; LS mean difference = -47.35, 90% CI 2-sided [-62.23 to -32.47], Standard Error of Mean 9.008 — Test group: PF-04965842 200 mg QD, Reference group: Placebo

3. Secondary Outcome: Percentage of Participants Achieving the IGA for Clear (0) or Almost Clear (1) and >=2 Points Improvement From Baseline at All Scheduled Time Points Except Week 12
Description: The IGA score quantifies the severity of participants' AD. Scores range from 0 to 4 and correspond to a category (clear, almost clear, mild, moderate and severe, respectively).
Time Frame: Baseline and all scheduled time points except Week 12, including Weeks 1, 2, 4, 6, 8, 13, 14, 16.
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | PF-04965842 10mg QD | PF-04965842 30mg QD | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 56 | 49 | 51 | 56 | 55
percentage of participants
  Week 1: number analyzed (Participants) | 54 | 48 | 50 | 55 | 54
  Week 1 | 0.0 | 2.1 | 2.0 | 1.8 | 3.7
  Week 2: number analyzed (Participants) | 55 | 49 | 50 | 55 | 52
  Week 2 | 3.6 | 6.1 | 6.0 | 3.6 | 11.5
  Week 4: number analyzed (Participants) | 55 | 49 | 50 | 55 | 54
  Week 4 | 1.8 | 8.2 | 8.0 | 16.4 | 40.7
  Week 6: number analyzed (Participants) | 55 | 49 | 50 | 55 | 54
  Week 6 | 14.5 | 14.3 | 14.0 | 12.7 | 40.7
  Week 8: number analyzed (Participants) | 55 | 49 | 50 | 55 | 53
  Week 8 | 5.5 | 8.2 | 12.0 | 16.4 | 41.5
  Week 13: number analyzed (Participants) | 30 | 29 | 31 | 38 | 45
  Week 13 | 10.0 | 20.7 | 12.9 | 23.7 | 26.7
  Week 14: number analyzed (Participants) | 32 | 28 | 29 | 40 | 44
  Week 14 | 18.8 | 10.7 | 3.4 | 12.5 | 15.9
  Week 16: number analyzed (Participants) | 28 | 26 | 27 | 36 | 38
  Week 16 | 10.7 | 23.1 | 7.4 | 13.9 | 18.4

4. Secondary Outcome: Percentage of Participants Achieving >=2 Points Improvement in the IGA From Baseline at All Scheduled Time Points
Description: as for outcome 3
Time Frame: Baseline and all scheduled time points, including Weeks 1, 2, 4, 6, 8, 12, 13, 14, 16
Population: "Number of Participants Analyzed" represents the number of participants in the FAS population. "Number Analyzed" at each visit represents the number of evaluable subjects for that visit.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | PF-04965842 10mg QD | PF-04965842 30mg QD | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 56 | 49 | 51 | 56 | 55
percentage of participants
  Week 1: number analyzed (Participants) | 54 | 48 | 49 | 55 | 53
  Week 1 | 1.9 | 4.2 | 6.1 | 5.5 | 9.4
  Week 2: number analyzed (Participants) | 55 | 48 | 47 | 53 | 50
  Week 2 | 7.3 | 10.4 | 10.6 | 11.3 | 24.0
  Week 4: number analyzed (Participants) | 50 | 45 | 47 | 52 | 52
  Week 4 | 8.0 | 11.1 | 12.8 | 25.0 | 51.9
  Week 6: number analyzed (Participants) | 44 | 38 | 43 | 48 | 52
  Week 6 | 22.7 | 23.7 | 18.6 | 29.2 | 59.6
  Week 8: number analyzed (Participants) | 41 | 36 | 43 | 47 | 49
  Week 8 | 14.6 | 19.4 | 23.3 | 34.0 | 59.2
  Week 12: number analyzed (Participants) | 35 | 29 | 30 | 43 | 42
  Week 12 | 17.1 | 17.2 | 23.3 | 51.2 | 57.1
  Week 13: number analyzed (Participants) | 30 | 29 | 31 | 38 | 45
  Week 13 | 13.3 | 24.1 | 12.9 | 26.3 | 37.8
  Week 14: number analyzed (Participants) | 32 | 28 | 29 | 40 | 44
  Week 14 | 21.9 | 17.9 | 10.3 | 20.0 | 25.0
  Week 16: number analyzed (Participants) | 28 | 26 | 27 | 36 | 38
  Week 16 | 14.3 | 26.9 | 11.1 | 22.2 | 31.6

5. Secondary Outcome: Percent Change From Baseline in the EASI Total Score at All Scheduled Time Points Except Week 12.
Description: The EASI quantifies the severity of participants' AD based on both severity of lesion clinical signs and the percent of BSA affected. EASI is a composite scoring by the AD clinical evaluator of the degree of erythema, induration/population, excoriation, and lichenification (each scored separately) for each of 4 regions, with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The EASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of AD.
Time Frame: Baseline and all scheduled time points except Week 12, including Weeks 1, 2, 4, 6, 8, 13, 14, 16
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | PF-04965842 10mg QD | PF-04965842 30mg QD | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 56 | 49 | 51 | 56 | 55
Percent change
  Week 1: number analyzed (Participants) | 54 | 48 | 49 | 55 | 53
  Week 1 | -12.28 (27.205) | -13.80 (26.526) | -14.85 (33.721) | -19.85 (30.379) | -41.26 (32.064)
  Week 2: number analyzed (Participants) | 55 | 48 | 47 | 53 | 50
  Week 2 | -23.54 (33.348) | -14.79 (40.474) | -26.29 (33.298) | -38.26 (39.176) | -63.28 (25.754)
  Week 4: number analyzed (Participants) | 50 | 45 | 47 | 52 | 52
  Week 4 | -24.58 (40.520) | -30.06 (40.852) | -32.81 (40.255) | -53.59 (35.274) | -78.16 (20.666)
  Week 6: number analyzed (Participants) | 44 | 38 | 43 | 48 | 52
  Week 6 | -39.17 (39.299) | -35.18 (43.498) | -40.16 (43.849) | -54.16 (53.212) | -83.14 (17.267)
  Week 8: number analyzed (Participants) | 41 | 36 | 43 | 47 | 49
  Week 8 | -36.69 (42.629) | -39.43 (46.270) | -36.83 (52.632) | -53.96 (53.689) | -84.48 (16.226)
  Week 13: number analyzed (Participants) | 30 | 29 | 31 | 38 | 45
  Week 13 | -29.82 (50.404) | -34.11 (51.089) | -32.97 (45.223) | -51.23 (45.968) | -66.34 (34.951)
  Week 14: number analyzed (Participants) | 32 | 28 | 29 | 40 | 44
  Week 14 | -35.51 (43.357) | -31.54 (62.829) | -26.25 (49.184) | -38.80 (49.085) | -57.15 (36.739)
  Week 16: number analyzed (Participants) | 28 | 26 | 27 | 36 | 38
  Week 16 | -35.91 (47.713) | -45.24 (44.576) | -20.80 (47.915) | -27.66 (54.570) | -55.82 (32.833)

6. Secondary Outcome: Percentage of Participants Achieving >=3 Points Improvement in the Pruritus Numerical Rating Scale (NRS) From Baseline at All Scheduled Time Points
Description: The severity of itch (pruritus) due to AD was assessed using a horizontal NRS. Participants were asked to assess their "worst itching due to AD over the past 24 hours" on a NRS anchored by the terms "no itching" (0) and "worst possible itching" (10).
  The frequency of itch (pruritus) due to AD was assessed using a horizontal NRS. Participants were asked to assess their "frequency of itching due to AD over the past 24 hours" on a NRS anchored by the terms "never/no itching" (0) and "always/constant itching" (10).
Time Frame: Baseline and all scheduled time points, including Days 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 29, 43, 57, 85, 99, 113
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | PF-04965842 10mg QD | PF-04965842 30mg QD | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 56 | 49 | 51 | 56 | 55
percentage of participants
  Itching due to AD Day 2: number analyzed (Participants) | 50 | 45 | 47 | 54 | 53
  Itching due to AD Day 2 | 4.0 | 6.7 | 17.0 | 14.8 | 17.0
  Itching due to AD Day 3: number analyzed (Participants) | 50 | 45 | 47 | 54 | 53
  Itching due to AD Day 3 | 8.0 | 2.2 | 14.9 | 22.2 | 28.3
  Itching due to AD Day 4: number analyzed (Participants) | 50 | 45 | 47 | 54 | 52
  Itching due to AD Day 4 | 2.0 | 2.2 | 21.3 | 22.2 | 34.6
  Itching due to AD Day 5: number analyzed (Participants) | 50 | 45 | 47 | 54 | 52
  Itching due to AD Day 5 | 2.0 | 6.7 | 29.8 | 24.1 | 36.5
  Itching due to AD Day 6: number analyzed (Participants) | 50 | 45 | 47 | 54 | 52
  Itching due to AD Day 6 | 10.0 | 8.9 | 25.5 | 24.1 | 40.4
  Itching due to AD Day 7: number analyzed (Participants) | 51 | 45 | 47 | 53 | 52
  Itching due to AD Day 7 | 11.8 | 13.3 | 25.5 | 30.2 | 42.3
  Itching due to AD Day 8: number analyzed (Participants) | 50 | 45 | 48 | 55 | 51
  Itching due to AD Day 8 | 10.0 | 13.3 | 25.0 | 43.6 | 51.0
  Itching due to AD Day 9: number analyzed (Participants) | 48 | 45 | 46 | 55 | 52
  Itching due to AD Day 9 | 8.3 | 11.1 | 26.1 | 45.5 | 50.0
  Itching due to AD Day 10: number analyzed (Participants) | 49 | 45 | 47 | 55 | 52
  Itching due to AD Day 10 | 8.2 | 11.1 | 34.0 | 43.6 | 55.8
  Itching due to AD Day 11: number analyzed (Participants) | 50 | 45 | 47 | 55 | 52
  Itching due to AD Day 11 | 16.0 | 15.6 | 27.7 | 43.6 | 57.7
  Itching due to AD Day 12: number analyzed (Participants) | 50 | 45 | 47 | 55 | 51
  Itching due to AD Day 12 | 22.0 | 17.8 | 38.3 | 49.1 | 60.8
  Itching due to AD Day 13: number analyzed (Participants) | 50 | 45 | 46 | 52 | 50
  Itching due to AD Day 13 | 24.0 | 15.6 | 28.3 | 53.8 | 66.0
  Itching due to AD Day 14: number analyzed (Participants) | 49 | 42 | 45 | 52 | 49
  Itching due to AD Day 14 | 22.4 | 19.0 | 26.7 | 48.1 | 67.3
  Itching due to AD Day 15: number analyzed (Participants) | 40 | 39 | 39 | 44 | 40
  Itching due to AD Day 15 | 25.0 | 17.9 | 30.8 | 54.5 | 72.5
  Itching due to AD Day 29: number analyzed (Participants) | 52 | 45 | 45 | 55 | 51
  Itching due to AD Day 29 | 32.7 | 31.1 | 37.8 | 60.0 | 74.5
  Itching due to AD Day 43: number analyzed (Participants) | 51 | 48 | 47 | 54 | 52
  Itching due to AD Day 43 | 31.4 | 35.4 | 38.3 | 53.7 | 73.1
  Itching due to AD Day 57: number analyzed (Participants) | 52 | 47 | 47 | 55 | 50
  Itching due to AD Day 57 | 28.8 | 31.9 | 38.3 | 54.5 | 72.0
  Itching due to AD Day 85: number analyzed (Participants) | 52 | 47 | 46 | 54 | 50
  Itching due to AD Day 85 | 26.9 | 21.3 | 41.3 | 53.7 | 64.0
  Itching due to AD Day 99: number analyzed (Participants) | 30 | 27 | 27 | 40 | 41
  Itching due to AD Day 99 | 33.3 | 25.9 | 33.3 | 47.5 | 41.5
  Itching due to AD Day 113: number analyzed (Participants) | 23 | 24 | 25 | 36 | 34
  Itching due to AD Day 113 | 52.2 | 29.2 | 24.0 | 44.4 | 35.3
  Frequency of itching due to AD Day 2: number analyzed (Participants) | 50 | 45 | 47 | 54 | 53
  Frequency of itching due to AD Day 2 | 6.0 | 8.9 | 19.1 | 22.2 | 26.4
  Frequency of itching due to AD Day 3: number analyzed (Participants) | 50 | 45 | 47 | 54 | 53
  Frequency of itching due to AD Day 3 | 10.0 | 8.9 | 19.1 | 25.9 | 34.0
  Frequency of itching due to AD Day 4: number analyzed (Participants) | 50 | 45 | 47 | 54 | 52
  Frequency of itching due to AD Day 4 | 8.0 | 4.4 | 23.4 | 25.9 | 48.1
  Frequency of itching due to AD Day 5: number analyzed (Participants) | 50 | 45 | 47 | 54 | 52
  Frequency of itching due to AD Day 5 | 10.0 | 6.7 | 31.9 | 29.6 | 46.2
  Frequency of itching due to AD Day 6: number analyzed (Participants) | 50 | 45 | 47 | 54 | 52
  Frequency of itching due to AD Day 6 | 14.0 | 8.9 | 27.7 | 33.3 | 57.7
  Frequency of itching due to AD Day 7: number analyzed (Participants) | 51 | 45 | 47 | 53 | 52
  Frequency of itching due to AD Day 7 | 15.7 | 11.1 | 31.9 | 34.0 | 55.8
  Frequency of itching due to AD Day 8: number analyzed (Participants) | 50 | 45 | 48 | 55 | 51
  Frequency of itching due to AD Day 8 | 16.0 | 11.1 | 29.2 | 45.5 | 60.8
  Frequency of itching due to AD Day 9: number analyzed (Participants) | 48 | 45 | 46 | 55 | 52
  Frequency of itching due to AD Day 9 | 14.6 | 13.3 | 30.4 | 45.5 | 55.8
  Frequency of itching due to AD Day 10: number analyzed (Participants) | 49 | 45 | 47 | 55 | 52
  Frequency of itching due to AD Day 10 | 14.3 | 13.3 | 36.2 | 45.5 | 65.4
  Frequency of itching due to AD Day 11: number analyzed (Participants) | 50 | 45 | 47 | 55 | 52
  Frequency of itching due to AD Day 11 | 20.0 | 15.6 | 36.2 | 45.5 | 63.5
  Frequency of itching due to AD Day 12: number analyzed (Participants) | 50 | 45 | 47 | 55 | 51
  Frequency of itching due to AD Day 12 | 18.0 | 17.8 | 38.3 | 50.9 | 60.8
  Frequency of itching due to AD Day 13: number analyzed (Participants) | 50 | 45 | 46 | 52 | 50
  Frequency of itching due to AD Day 13 | 20.0 | 20.0 | 30.4 | 51.9 | 70.0
  Frequency of itching due to AD Day 14: number analyzed (Participants) | 49 | 42 | 45 | 52 | 49
  Frequency of itching due to AD Day 14 | 24.5 | 23.8 | 33.3 | 48.1 | 71.4
  Frequency of itching due to AD Day 15: number analyzed (Participants) | 40 | 39 | 39 | 44 | 40
  Frequency of itching due to AD Day 15 | 30.0 | 20.5 | 38.5 | 52.3 | 72.5
  Frequency of itching due to AD Day 29: number analyzed (Participants) | 52 | 45 | 45 | 55 | 51
  Frequency of itching due to AD Day 29 | 28.8 | 28.9 | 40.0 | 60.0 | 74.5
  Frequency of itching due to AD Day 43: number analyzed (Participants) | 51 | 48 | 47 | 54 | 52
  Frequency of itching due to AD Day 43 | 23.5 | 35.4 | 38.3 | 57.4 | 75.0
  Frequency of itching due to AD Day 57: number analyzed (Participants) | 52 | 47 | 47 | 55 | 50
  Frequency of itching due to AD Day 57 | 26.9 | 29.8 | 38.3 | 54.5 | 74.0
  Frequency of itching due to AD Day 85: number analyzed (Participants) | 52 | 47 | 46 | 54 | 50
  Frequency of itching due to AD Day 85 | 25.0 | 25.5 | 34.8 | 53.7 | 70.0
  Frequency of itching due to AD Day 99: number analyzed (Participants) | 30 | 27 | 27 | 40 | 41
  Frequency of itching due to AD Day 99 | 30.0 | 22.2 | 37.0 | 47.5 | 39.0
  Frequency of itching due to AD Day 113: number analyzed (Participants) | 23 | 24 | 25 | 36 | 34
  Frequency of itching due to AD Day 113 | 47.8 | 25.0 | 20.0 | 47.2 | 38.2

7. Secondary Outcome: Percentage of Participants Achieving >=4 Points Improvement in the Pruritus NRS From Baseline at All Scheduled Time Points
Description: as for outcome 6
Time Frame: as for outcome 6
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | PF-04965842 10mg QD | PF-04965842 30mg QD | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 56 | 49 | 51 | 56 | 55
percentage of participants
  Itching due to AD Day 2: number analyzed (Participants) | 49 | 45 | 46 | 50 | 46
  Itching due to AD Day 2 | 2.0 | 2.2 | 6.5 | 10.0 | 15.2
  Itching due to AD Day 3: number analyzed (Participants) | 49 | 45 | 46 | 50 | 46
  Itching due to AD Day 3 | 0.0 | 2.2 | 13.0 | 14.0 | 21.7
  Itching due to AD Day 4: number analyzed (Participants) | 49 | 45 | 46 | 50 | 45
  Itching due to AD Day 4 | 0.0 | 0.0 | 17.4 | 14.0 | 28.9
  Itching due to AD Day 5: number analyzed (Participants) | 49 | 45 | 46 | 50 | 45
  Itching due to AD Day 5 | 2.0 | 2.2 | 19.6 | 20.0 | 26.7
  Itching due to AD Day 6: number analyzed (Participants) | 49 | 45 | 46 | 50 | 45
  Itching due to AD Day 6 | 6.1 | 2.2 | 17.4 | 24.0 | 35.6
  Itching due to AD Day 7: number analyzed (Participants) | 50 | 45 | 46 | 49 | 45
  Itching due to AD Day 7 | 8.0 | 8.9 | 19.6 | 20.4 | 37.8
  Itching due to AD Day 8: number analyzed (Participants) | 49 | 45 | 47 | 51 | 44
  Itching due to AD Day 8 | 6.1 | 4.4 | 14.9 | 29.4 | 52.3
  Itching due to AD Day 9: number analyzed (Participants) | 47 | 45 | 45 | 51 | 45
  Itching due to AD Day 9 | 2.1 | 6.7 | 20.0 | 27.5 | 51.1
  Itching due to AD Day 10: number analyzed (Participants) | 48 | 45 | 46 | 51 | 45
  Itching due to AD Day 10 | 4.2 | 6.7 | 21.7 | 29.4 | 44.4
  Itching due to AD Day 11: number analyzed (Participants) | 49 | 45 | 46 | 51 | 45
  Itching due to AD Day 11 | 8.2 | 13.3 | 19.6 | 29.4 | 44.4
  Itching due to AD Day 12: number analyzed (Participants) | 49 | 45 | 46 | 51 | 45
  Itching due to AD Day 12 | 10.2 | 11.1 | 23.9 | 35.3 | 51.1
  Itching due to AD Day 13: number analyzed (Participants) | 49 | 45 | 45 | 49 | 44
  Itching due to AD Day 13 | 14.3 | 6.7 | 20.0 | 38.8 | 61.4
  Itching due to AD Day 14: number analyzed (Participants) | 48 | 42 | 44 | 48 | 44
  Itching due to AD Day 14 | 10.4 | 14.3 | 25.0 | 41.7 | 59.1
  Itching due to AD Day 15: number analyzed (Participants) | 40 | 38 | 38 | 43 | 37
  Itching due to AD Day 15 | 15.0 | 7.9 | 31.6 | 41.9 | 70.3
  Itching due to AD Day 29: number analyzed (Participants) | 51 | 44 | 44 | 51 | 45
  Itching due to AD Day 29 | 17.6 | 13.6 | 25.0 | 52.9 | 68.9
  Itching due to AD Day 43: number analyzed (Participants) | 50 | 45 | 46 | 50 | 46
  Itching due to AD Day 43 | 20.0 | 22.2 | 23.9 | 50.0 | 71.7
  Itching due to AD Day 57: number analyzed (Participants) | 51 | 44 | 46 | 51 | 44
  Itching due to AD Day 57 | 17.6 | 22.7 | 26.1 | 52.9 | 72.7
  Itching due to AD Day 85: number analyzed (Participants) | 51 | 44 | 45 | 50 | 44
  Itching due to AD Day 85 | 25.5 | 22.7 | 33.3 | 50.0 | 63.6
  Itching due to AD Day 99: number analyzed (Participants) | 29 | 27 | 26 | 39 | 35
  Itching due to AD Day 99 | 27.6 | 25.9 | 23.1 | 38.5 | 37.1
  Itching due to AD Day 113: number analyzed (Participants) | 23 | 24 | 24 | 35 | 29
  Itching due to AD Day 113 | 43.5 | 20.8 | 16.7 | 34.3 | 31.0
  Frequency of itching due to AD Day 2: number analyzed (Participants) | 47 | 45 | 42 | 52 | 48
  Frequency of itching due to AD Day 2 | 2.1 | 0.0 | 7.1 | 11.5 | 18.8
  Frequency of itching due to AD Day 3: number analyzed (Participants) | 47 | 45 | 42 | 52 | 48
  Frequency of itching due to AD Day 3 | 6.4 | 2.2 | 11.9 | 13.5 | 22.9
  Frequency of itching due to AD Day 4: number analyzed (Participants) | 47 | 45 | 42 | 52 | 47
  Frequency of itching due to AD Day 4 | 2.1 | 0.0 | 19.0 | 21.2 | 36.2
  Frequency of itching due to AD Day 5: number analyzed (Participants) | 47 | 45 | 42 | 52 | 47
  Frequency of itching due to AD Day 5 | 4.3 | 4.4 | 23.8 | 25.0 | 38.3
  Frequency of itching due to AD Day 6: number analyzed (Participants) | 47 | 45 | 42 | 52 | 47
  Frequency of itching due to AD Day 6 | 10.6 | 6.7 | 26.2 | 25.0 | 44.7
  Frequency of itching due to AD Day 7: number analyzed (Participants) | 48 | 45 | 42 | 50 | 47
  Frequency of itching due to AD Day 7 | 10.4 | 4.4 | 19.0 | 30.0 | 51.1
  Frequency of itching due to AD Day 8: number analyzed (Participants) | 47 | 45 | 43 | 52 | 46
  Frequency of itching due to AD Day 8 | 8.5 | 2.2 | 23.3 | 36.5 | 54.3
  Frequency of itching due to AD Day 9: number analyzed (Participants) | 45 | 45 | 41 | 52 | 47
  Frequency of itching due to AD Day 9 | 6.7 | 6.7 | 26.8 | 36.5 | 48.9
  Frequency of itching due to AD Day 10: number analyzed (Participants) | 46 | 45 | 42 | 52 | 47
  Frequency of itching due to AD Day 10 | 6.5 | 8.9 | 31.0 | 28.8 | 51.1
  Frequency of itching due to AD Day 11: number analyzed (Participants) | 47 | 45 | 42 | 52 | 47
  Frequency of itching due to AD Day 11 | 10.6 | 15.6 | 23.8 | 32.7 | 55.3
  Frequency of itching due to AD Day 12: number analyzed (Participants) | 47 | 45 | 42 | 52 | 46
  Frequency of itching due to AD Day 12 | 12.8 | 13.3 | 26.2 | 34.6 | 54.3
  Frequency of itching due to AD Day 13: number analyzed (Participants) | 47 | 45 | 41 | 50 | 45
  Frequency of itching due to AD Day 13 | 17.0 | 15.6 | 29.3 | 32.0 | 66.7
  Frequency of itching due to AD Day 14: number analyzed (Participants) | 46 | 42 | 40 | 49 | 45
  Frequency of itching due to AD Day 14 | 19.6 | 16.7 | 30.0 | 34.7 | 66.7
  Frequency of itching due to AD Day 15: number analyzed (Participants) | 40 | 38 | 34 | 44 | 38
  Frequency of itching due to AD Day 15 | 20.0 | 15.8 | 35.3 | 36.4 | 71.1
  Frequency of itching due to AD Day 29: number analyzed (Participants) | 49 | 44 | 40 | 52 | 47
  Frequency of itching due to AD Day 29 | 16.3 | 15.9 | 35.0 | 51.9 | 66.0
  Frequency of itching due to AD Day 43: number analyzed (Participants) | 48 | 45 | 42 | 51 | 48
  Frequency of itching due to AD Day 43 | 12.5 | 24.4 | 28.6 | 58.8 | 72.9
  Frequency of itching due to AD Day 57: number analyzed (Participants) | 49 | 44 | 42 | 52 | 46
  Frequency of itching due to AD Day 57 | 16.3 | 20.5 | 33.3 | 53.8 | 73.9
  Frequency of itching due to AD Day 85: number analyzed (Participants) | 49 | 44 | 42 | 51 | 46
  Frequency of itching due to AD Day 85 | 24.5 | 25.0 | 28.6 | 47.1 | 69.6
  Frequency of itching due to AD Day 99: number analyzed (Participants) | 29 | 27 | 24 | 38 | 37
  Frequency of itching due to AD Day 99 | 20.7 | 18.5 | 16.7 | 39.5 | 32.4
  Frequency of itching due to AD Day 113: number analyzed (Participants) | 23 | 24 | 22 | 34 | 30
  Frequency of itching due to AD Day 113 | 34.8 | 20.8 | 22.7 | 29.4 | 26.7

8. Secondary Outcome: Time to Achieving >=3 Points Improvement in NRS
Description: as for outcome 6
Time Frame: Baseline till Week 16
Population: as for outcome 4
Measure: Median (90% Confidence Interval); unit: day
Arm/Group | Placebo | PF-04965842 10mg QD | PF-04965842 30mg QD | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 56 | 49 | 51 | 56 | 55
day
  Itching due to AD: number analyzed (Participants) | 55 | 49 | 50 | 55 | 54
  Itching due to AD | 30.0 [15.0 to 56.0] | 43.0 [29.0 to 57.0] | 12.0 [8.0 to 30.0] | 9.0 [7.0 to 14.0] | 7.0 [5.0 to 11.0]
  Frequency of itching due to AD: number analyzed (Participants) | 55 | 49 | 50 | 55 | 54
  Frequency of itching due to AD | 29.0 [13.0 to 57.0] | 43.0 [29.0 to 85.0] | 13.0 [7.0 to 43.0] | 8.0 [4.0 to 10.0] | 4.0 [4.0 to 6.0]

9. Secondary Outcome: Time to Achieving >=4 Points Improvement in NRS
Description: as for outcome 6
Time Frame: Baseline till Week 16
Population: as for outcome 4
Measure: Median (90% Confidence Interval); unit: day
Arm/Group | Placebo | PF-04965842 10mg QD | PF-04965842 30mg QD | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 56 | 49 | 51 | 56 | 55
day
  Itching due to atopic dermatitis: number analyzed (Participants) | 55 | 49 | 50 | 55 | 54
  Itching due to atopic dermatitis | 78.0 [56.0 to NA] — The NA was generated because of the high censoring rates in the placebo group. | NA [47.0 to NA] — The NA was generated because of the high censoring rates in the PF-04965842 10 mg group. | 43.0 [15.0 to 85.0] | 14.0 [10.0 to 29.0] | 10.0 [7.0 to 13.0]
  Frequency of itching due to atopic dermatitis: number analyzed (Participants) | 55 | 49 | 50 | 55 | 54
  Frequency of itching due to atopic dermatitis | 59.0 [30.0 to NA] — The NA was generated because of the high censoring rates in the placebo group. | NA [56.0 to NA] — The NA was generated because of the high censoring rates in the PF-04965842 10 mg group. | 29.0 [12.0 to 98.0] | 14.0 [8.0 to 29.0] | 7.0 [5.0 to 9.0]

10. Secondary Outcome: Percent Change From Baseline in the Pruritus NRS From Baseline at All Scheduled Time Points
Description: as for outcome 6
Time Frame: as for outcome 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04965842 10mg QD | PF-04965842 30mg QD | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 56 | 49 | 51 | 56 | 55
percent change
  Itching due to AD Day 2: number analyzed (Participants) | 50 | 45 | 47 | 53 | 51
  Itching due to AD Day 2 | 0.56 (19.298) | -1.51 (19.857) | -9.39 (23.528) | -10.06 (25.930) | -6.79 (47.751)
  Itching due to AD Day 3: number analyzed (Participants) | 50 | 45 | 47 | 52 | 51
  Itching due to AD Day 3 | -1.32 (22.630) | 2.48 (21.994) | -8.22 (33.257) | -15.32 (27.874) | -16.72 (40.055)
  Itching due to AD Day 4: number analyzed (Participants) | 50 | 44 | 47 | 52 | 50
  Itching due to AD Day 4 | -1.98 (22.326) | 0.23 (17.314) | -12.18 (33.385) | -17.62 (25.747) | -25.80 (38.557)
  Itching due to AD Day 5: number analyzed (Participants) | 50 | 44 | 47 | 52 | 50
  Itching due to AD Day 5 | -2.98 (22.385) | -2.37 (20.174) | -18.92 (31.846) | -20.48 (27.983) | -30.91 (34.215)
  Itching due to AD Day 6: number analyzed (Participants) | 50 | 44 | 47 | 52 | 50
  Itching due to AD Day 6 | -1.52 (25.690) | -5.70 (23.478) | -16.70 (33.407) | -21.58 (27.842) | -34.02 (35.532)
  Itching due to AD Day 7: number analyzed (Participants) | 51 | 44 | 47 | 51 | 50
  Itching due to AD Day 7 | -4.18 (30.531) | -4.59 (28.248) | -18.07 (33.640) | -23.02 (33.524) | -38.17 (35.428)
  Itching due to AD Day 8: number analyzed (Participants) | 50 | 44 | 46 | 53 | 49
  Itching due to AD Day 8 | -0.35 (34.144) | -5.69 (25.576) | -17.87 (34.789) | -32.36 (30.610) | -43.13 (38.684)
  Itching due to AD Day 9: number analyzed (Participants) | 48 | 44 | 42 | 51 | 49
  Itching due to AD Day 9 | -2.56 (30.688) | -8.61 (27.803) | -22.74 (33.667) | -31.82 (30.951) | -39.37 (41.055)
  Itching due to AD Day 10: number analyzed (Participants) | 49 | 44 | 43 | 51 | 49
  Itching due to AD Day 10 | -3.32 (29.885) | -5.97 (29.093) | -22.90 (41.573) | -31.93 (27.094) | -39.60 (56.607)
  Itching due to AD Day 11: number analyzed (Participants) | 49 | 44 | 43 | 51 | 49
  Itching due to AD Day 11 | -7.81 (30.201) | -5.94 (31.028) | -16.76 (49.412) | -33.13 (27.902) | -42.50 (51.621)
  Itching due to AD Day 12: number analyzed (Participants) | 49 | 44 | 43 | 51 | 48
  Itching due to AD Day 12 | -11.12 (30.087) | -6.65 (32.617) | -27.84 (33.416) | -33.30 (34.252) | -46.40 (46.241)
  Itching due to AD Day 13: number analyzed (Participants) | 48 | 44 | 42 | 49 | 47
  Itching due to AD Day 13 | -15.16 (29.759) | -7.43 (27.374) | -24.56 (30.086) | -35.89 (35.651) | -49.77 (48.426)
  Itching due to AD Day 14: number analyzed (Participants) | 47 | 41 | 41 | 48 | 46
  Itching due to AD Day 14 | -13.61 (30.153) | -8.84 (29.474) | -26.70 (29.805) | -36.57 (27.552) | -55.45 (34.331)
  Itching due to AD Day 15: number analyzed (Participants) | 38 | 35 | 35 | 42 | 38
  Itching due to AD Day 15 | -17.24 (30.755) | -7.28 (28.058) | -25.09 (37.815) | -35.41 (29.140) | -59.00 (39.804)
  Itching due to AD Day 29: number analyzed (Participants) | 46 | 41 | 41 | 51 | 49
  Itching due to AD Day 29 | -19.43 (35.575) | -16.63 (34.554) | -28.41 (36.183) | -46.62 (40.090) | -68.09 (31.214)
  Itching due to AD Day 43: number analyzed (Participants) | 40 | 37 | 40 | 46 | 50
  Itching due to AD Day 43 | -26.55 (36.418) | -27.15 (39.550) | -31.14 (39.090) | -49.49 (46.279) | -67.80 (36.372)
  Itching due to AD Day 57: number analyzed (Participants) | 38 | 34 | 40 | 46 | 46
  Itching due to AD Day 57 | -25.54 (39.577) | -21.60 (44.446) | -29.60 (39.606) | -54.11 (36.374) | -70.13 (36.338)
  Itching due to AD Day 85: number analyzed (Participants) | 35 | 30 | 31 | 42 | 44
  Itching due to AD Day 85 | -30.10 (42.697) | -22.47 (48.291) | -30.39 (47.772) | -56.51 (41.955) | -53.66 (109.454)
  Itching due to AD Day 99: number analyzed (Participants) | 30 | 27 | 27 | 39 | 41
  Itching due to AD Day 99 | -19.24 (43.251) | -15.94 (42.332) | -11.46 (39.959) | -32.68 (34.789) | 5.61 (139.223)
  Itching due to AD Day 113: number analyzed (Participants) | 23 | 24 | 25 | 35 | 34
  Itching due to AD Day 113 | -31.99 (45.929) | -14.07 (47.186) | -14.34 (29.756) | -28.47 (41.027) | 24.61 (190.848)
  Frequency of itching due to AD Day 2: number analyzed (Participants) | 50 | 45 | 47 | 53 | 52
  Frequency of itching due to AD Day 2 | 6.72 (45.759) | -6.67 (19.016) | -10.14 (28.184) | -17.93 (20.967) | -10.52 (79.180)
  Frequency of itching due to AD Day 3: number analyzed (Participants) | 50 | 45 | 47 | 52 | 52
  Frequency of itching due to AD Day 3 | 2.59 (45.541) | 0.30 (24.330) | -3.96 (49.425) | -19.98 (22.910) | -16.46 (67.794)
  Frequency of itching due to AD Day 4: number analyzed (Participants) | 50 | 44 | 47 | 52 | 51
  Frequency of itching due to AD Day 4 | 3.73 (37.683) | -3.25 (15.230) | -9.39 (39.225) | -20.71 (24.391) | -28.27 (47.925)
  Frequency of itching due to AD Day 5: number analyzed (Participants) | 50 | 44 | 47 | 52 | 51
  Frequency of itching due to AD Day 5 | -0.70 (34.834) | -3.73 (23.125) | -17.72 (38.967) | -23.69 (24.954) | -35.45 (37.436)
  Frequency of itching due to AD Day 6: number analyzed (Participants) | 50 | 44 | 47 | 52 | 51
  Frequency of itching due to AD Day 6 | 4.04 (52.799) | -5.76 (24.623) | -14.84 (38.256) | -26.47 (27.218) | -44.31 (36.476)
  Frequency of itching due to AD Day 7: number analyzed (Participants) | 51 | 44 | 47 | 51 | 51
  Frequency of itching due to AD Day 7 | -2.25 (37.193) | -3.56 (25.414) | -17.05 (40.108) | -27.80 (32.466) | -40.19 (39.702)
  Frequency of itching due to AD Day 8: number analyzed (Participants) | 50 | 44 | 46 | 53 | 50
  Frequency of itching due to AD Day 8 | 1.22 (38.544) | -3.90 (25.515) | -19.05 (36.488) | -35.44 (29.791) | -46.26 (43.491)
  Frequency of itching due to AD Day 9: number analyzed (Participants) | 48 | 44 | 42 | 51 | 50
  Frequency of itching due to AD Day 9 | 1.08 (58.633) | -8.79 (26.589) | -17.58 (42.054) | -35.17 (29.637) | -44.29 (43.238)
  Frequency of itching due to AD Day 10: number analyzed (Participants) | 49 | 44 | 43 | 51 | 50
  Frequency of itching due to AD Day 10 | -3.47 (53.518) | -5.41 (32.491) | -19.84 (47.884) | -33.23 (26.950) | -49.78 (37.349)
  Frequency of itching due to AD Day 11: number analyzed (Participants) | 49 | 44 | 43 | 51 | 50
  Frequency of itching due to AD Day 11 | -6.24 (49.163) | -5.88 (32.750) | -18.73 (42.599) | -34.93 (27.181) | -51.62 (37.385)
  Frequency of itching due to AD Day 12: number analyzed (Participants) | 49 | 44 | 43 | 51 | 49
  Frequency of itching due to AD Day 12 | -8.41 (49.918) | -5.65 (36.637) | -25.00 (31.695) | -36.55 (27.281) | -51.92 (40.010)
  Frequency of itching due to AD Day 13: number analyzed (Participants) | 48 | 44 | 42 | 49 | 48
  Frequency of itching due to AD Day 13 | -13.45 (40.159) | -10.46 (31.103) | -24.73 (31.960) | -35.75 (32.757) | -53.17 (40.695)
  Frequency of itching due to AD Day 14: number analyzed (Participants) | 47 | 41 | 41 | 48 | 47
  Frequency of itching due to AD Day 14 | -10.26 (46.126) | -13.86 (32.390) | -27.70 (30.476) | -38.28 (27.724) | -57.50 (39.073)
  Frequency of itching due to AD Day 15: number analyzed (Participants) | 38 | 35 | 35 | 42 | 38
  Frequency of itching due to AD Day 15 | -18.78 (34.923) | -11.34 (28.494) | -26.88 (38.846) | -38.87 (29.184) | -60.99 (32.840)
  Frequency of itching due to AD Day 29: number analyzed (Participants) | 46 | 41 | 41 | 51 | 49
  Frequency of itching due to AD Day 29 | -16.05 (39.630) | -17.15 (33.432) | -28.55 (43.421) | -49.94 (36.649) | -67.84 (29.918)
  Frequency of itching due to AD Day 43: number analyzed (Participants) | 40 | 37 | 40 | 46 | 50
  Frequency of itching due to AD Day 43 | -24.51 (30.798) | -32.19 (37.806) | -26.48 (46.793) | -53.95 (41.772) | -69.24 (38.370)
  Frequency of itching due to AD Day 57: number analyzed (Participants) | 38 | 34 | 40 | 46 | 46
  Frequency of itching due to AD Day 57 | -24.94 (35.662) | -23.28 (44.257) | -27.91 (39.142) | -55.39 (35.447) | -73.50 (30.583)
  Frequency of itching due to AD Day 85: number analyzed (Participants) | 35 | 30 | 31 | 42 | 44
  Frequency of itching due to AD Day 85 | -29.81 (44.035) | -25.76 (43.273) | -32.28 (38.817) | -54.51 (43.354) | -54.54 (120.723)
  Frequency of itching due to AD Day 99: number analyzed (Participants) | 30 | 27 | 27 | 39 | 41
  Frequency of itching due to AD Day 99 | -17.46 (43.552) | -20.21 (36.947) | -3.36 (52.153) | -13.57 (123.800) | 2.12 (144.572)
  Frequency of itching due to AD Day 113: number analyzed (Participants) | 23 | 24 | 25 | 35 | 34
  Frequency of itching due to AD Day 113 | -28.95 (46.896) | -16.22 (38.055) | -5.65 (51.132) | -12.62 (113.423) | 27.77 (203.937)

11. Secondary Outcome: Change From Baseline in Pruritus NRS Score at All Scheduled Time Points
Description: as for outcome 6
Time Frame: as for outcome 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | PF-04965842 10mg QD | PF-04965842 30mg QD | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 56 | 49 | 51 | 56 | 55
units on a scale
  Itching due to AD Day 2: number analyzed (Participants) | 50 | 45 | 47 | 54 | 52
  Itching due to AD Day 2 | -0.08 (1.307) | -0.20 (1.217) | -0.83 (1.672) | -0.85 (1.607) | -1.00 (2.433)
  Itching due to AD Day 3: number analyzed (Participants) | 50 | 45 | 47 | 53 | 52
  Itching due to AD Day 3 | -0.22 (1.418) | 0.02 (1.357) | -0.85 (2.095) | -1.21 (1.702) | -1.48 (2.493)
  Itching due to AD Day 4: number analyzed (Participants) | 50 | 44 | 47 | 53 | 51
  Itching due to AD Day 4 | -0.22 (1.389) | -0.09 (1.117) | -1.09 (2.263) | -1.26 (1.862) | -2.12 (2.590)
  Itching due to AD Day 5: number analyzed (Participants) | 50 | 44 | 47 | 53 | 51
  Itching due to AD Day 5 | -0.32 (1.406) | -0.27 (1.264) | -1.55 (2.348) | -1.58 (1.865) | -2.35 (2.583)
  Itching due to AD Day 6: number analyzed (Participants) | 50 | 44 | 47 | 53 | 51
  Itching due to AD Day 6 | -0.28 (1.727) | -0.55 (1.405) | -1.47 (2.492) | -1.49 (2.317) | -2.53 (2.648)
  Itching due to AD Day 7: number analyzed (Participants) | 51 | 44 | 47 | 52 | 51
  Itching due to AD Day 7 | -0.53 (2.023) | -0.52 (1.745) | -1.51 (2.422) | -1.75 (2.159) | -2.77 (2.795)
  Itching due to AD Day 8: number analyzed (Participants) | 50 | 44 | 46 | 54 | 50
  Itching due to AD Day 8 | -0.30 (2.215) | -0.56 (1.560) | -1.65 (2.514) | -2.39 (2.294) | -3.22 (3.039)
  Itching due to AD Day 9: number analyzed (Participants) | 48 | 44 | 42 | 52 | 50
  Itching due to AD Day 9 | -0.38 (2.080) | -0.75 (1.844) | -1.95 (2.527) | -2.40 (2.154) | -3.18 (2.988)
  Itching due to AD Day 10: number analyzed (Participants) | 49 | 44 | 43 | 52 | 50
  Itching due to AD Day 10 | -0.43 (1.947) | -0.61 (1.967) | -2.09 (2.698) | -2.21 (2.412) | -3.38 (2.975)
  Itching due to AD Day 11: number analyzed (Participants) | 49 | 44 | 43 | 52 | 50
  Itching due to AD Day 11 | -0.73 (1.955) | -0.61 (2.148) | -1.72 (2.462) | -2.33 (2.415) | -3.40 (3.071)
  Itching due to AD Day 12: number analyzed (Participants) | 49 | 44 | 43 | 52 | 49
  Itching due to AD Day 12 | -0.92 (1.988) | -0.73 (2.245) | -2.28 (2.271) | -2.46 (2.578) | -3.63 (3.154)
  Itching due to AD Day 13: number analyzed (Participants) | 48 | 44 | 42 | 49 | 48
  Itching due to AD Day 13 | -1.21 (1.989) | -0.68 (1.801) | -1.98 (2.268) | -2.84 (2.164) | -3.88 (3.085)
  Itching due to AD Day 14: number analyzed (Participants) | 47 | 41 | 41 | 49 | 47
  Itching due to AD Day 14 | -1.11 (2.003) | -0.78 (2.104) | -2.10 (2.211) | -2.53 (2.567) | -4.06 (2.793)
  Itching due to AD Day 15: number analyzed (Participants) | 38 | 35 | 35 | 42 | 38
  Itching due to AD Day 15 | -1.39 (2.034) | -0.69 (1.937) | -2.06 (2.508) | -2.79 (2.290) | -4.37 (2.696)
  Itching due to AD Day 29: number analyzed (Participants) | 46 | 41 | 41 | 52 | 49
  Itching due to AD Day 29 | -1.63 (2.453) | -1.34 (2.383) | -2.17 (2.519) | -3.58 (3.322) | -5.00 (2.880)
  Itching due to AD Day 43: number analyzed (Participants) | 40 | 37 | 40 | 47 | 50
  Itching due to AD Day 43 | -1.93 (2.325) | -2.24 (2.929) | -2.50 (2.562) | -3.77 (3.778) | -5.02 (3.172)
  Itching due to AD Day 57: number analyzed (Participants) | 38 | 34 | 40 | 47 | 46
  Itching due to AD Day 57 | -1.84 (2.594) | -1.97 (3.398) | -2.55 (2.943) | -4.00 (3.336) | -5.26 (3.130)
  Itching due to AD Day 85: number analyzed (Participants) | 35 | 30 | 31 | 43 | 44
  Itching due to AD Day 85 | -2.26 (3.081) | -2.13 (3.711) | -2.68 (2.749) | -4.21 (3.529) | -4.84 (3.785)
  Itching due to AD Day 99: number analyzed (Participants) | 30 | 27 | 27 | 40 | 41
  Itching due to AD Day 99 | -1.57 (3.025) | -1.48 (2.992) | -1.37 (2.452) | -2.28 (2.900) | -1.90 (3.767)
  Itching due to AD Day 113: number analyzed (Participants) | 23 | 24 | 25 | 36 | 34
  Itching due to AD Day 113 | -2.43 (3.259) | -1.38 (3.201) | -1.32 (2.410) | -2.03 (3.185) | -1.50 (3.736)
  Frequency of itching due to AD Day 2: number analyzed (Participants) | 50 | 45 | 47 | 54 | 52
  Frequency of itching due to AD Day 2 | -0.06 (1.754) | -0.44 (1.198) | -0.94 (1.737) | -1.35 (1.556) | -1.60 (2.345)
  Frequency of itching due to AD Day 3: number analyzed (Participants) | 50 | 45 | 47 | 53 | 52
  Frequency of itching due to AD Day 3 | -0.38 (1.894) | -0.16 (1.461) | -0.79 (2.331) | -1.49 (1.694) | -1.92 (2.300)
  Frequency of itching due to AD Day 4: number analyzed (Participants) | 50 | 44 | 47 | 53 | 51
  Frequency of itching due to AD Day 4 | -0.20 (1.738) | -0.32 (1.073) | -1.02 (2.162) | -1.40 (2.069) | -2.47 (2.533)
  Frequency of itching due to AD Day 5: number analyzed (Participants) | 50 | 44 | 47 | 53 | 51
  Frequency of itching due to AD Day 5 | -0.42 (1.727) | -0.43 (1.516) | -1.49 (2.349) | -1.75 (1.828) | -2.73 (2.515)
  Frequency of itching due to AD Day 6: number analyzed (Participants) | 50 | 44 | 47 | 53 | 51
  Frequency of itching due to AD Day 6 | -0.40 (2.250) | -0.55 (1.606) | -1.40 (2.402) | -1.77 (2.326) | -3.24 (2.446)
  Frequency of itching due to AD Day 7: number analyzed (Participants) | 51 | 44 | 47 | 52 | 51
  Frequency of itching due to AD Day 7 | -0.63 (2.181) | -0.43 (1.676) | -1.53 (2.466) | -2.04 (2.214) | -3.15 (2.739)
  Frequency of itching due to AD Day 8: number analyzed (Participants) | 50 | 44 | 46 | 54 | 50
  Frequency of itching due to AD Day 8 | -0.42 (2.205) | -0.40 (1.679) | -1.74 (2.542) | -2.59 (2.278) | -3.69 (2.808)
  Frequency of itching due to AD Day 9: number analyzed (Participants) | 48 | 44 | 42 | 52 | 50
  Frequency of itching due to AD Day 9 | -0.54 (2.240) | -0.75 (2.036) | -1.74 (2.567) | -2.62 (2.268) | -3.54 (3.018)
  Frequency of itching due to AD Day 10: number analyzed (Participants) | 49 | 44 | 43 | 52 | 50
  Frequency of itching due to AD Day 10 | -0.80 (2.198) | -0.64 (2.200) | -1.84 (2.760) | -2.33 (2.565) | -3.68 (2.591)
  Frequency of itching due to AD Day 11: number analyzed (Participants) | 49 | 44 | 43 | 52 | 50
  Frequency of itching due to AD Day 11 | -0.96 (2.336) | -0.68 (2.380) | -1.79 (2.541) | -2.46 (2.540) | -3.74 (2.633)
  Frequency of itching due to AD Day 12: number analyzed (Participants) | 49 | 44 | 43 | 52 | 49
  Frequency of itching due to AD Day 12 | -1.06 (2.322) | -0.66 (2.411) | -2.00 (2.182) | -2.54 (2.509) | -3.84 (2.932)
  Frequency of itching due to AD Day 13: number analyzed (Participants) | 48 | 44 | 42 | 49 | 48
  Frequency of itching due to AD Day 13 | -1.33 (2.337) | -0.91 (2.133) | -1.90 (2.195) | -2.78 (2.275) | -4.08 (2.952)
  Frequency of itching due to AD Day 14: number analyzed (Participants) | 47 | 41 | 41 | 49 | 47
  Frequency of itching due to AD Day 14 | -1.17 (2.417) | -1.10 (2.417) | -2.00 (2.225) | -2.63 (2.620) | -4.28 (2.841)
  Frequency of itching due to AD Day 15: number analyzed (Participants) | 38 | 35 | 35 | 42 | 38
  Frequency of itching due to AD Day 15 | -1.50 (2.322) | -0.97 (2.135) | -2.17 (2.407) | -3.02 (2.464) | -4.50 (2.648)
  Frequency of itching due to AD Day 29: number analyzed (Participants) | 46 | 41 | 41 | 52 | 49
  Frequency of itching due to AD Day 29 | -1.46 (2.518) | -1.34 (2.425) | -2.22 (2.761) | -3.77 (3.317) | -5.06 (2.817)
  Frequency of itching due to AD Day 43: number analyzed (Participants) | 40 | 37 | 40 | 47 | 50
  Frequency of itching due to AD Day 43 | -1.70 (1.990) | -2.51 (3.061) | -2.28 (2.953) | -4.02 (3.796) | -5.30 (2.957)
  Frequency of itching due to AD Day 57: number analyzed (Participants) | 38 | 34 | 40 | 47 | 46
  Frequency of itching due to AD Day 57 | -1.74 (2.298) | -2.00 (3.499) | -2.45 (2.943) | -4.02 (3.467) | -5.59 (3.037)
  Frequency of itching due to AD Day 85: number analyzed (Participants) | 35 | 30 | 31 | 43 | 44
  Frequency of itching due to AD Day 85 | -2.23 (3.209) | -2.33 (3.575) | -2.61 (2.692) | -4.09 (3.663) | -5.14 (3.645)
  Frequency of itching due to AD Day 99: number analyzed (Participants) | 30 | 27 | 27 | 40 | 41
  Frequency of itching due to AD Day 99 | -1.30 (2.781) | -1.56 (2.736) | -0.93 (2.526) | -2.03 (3.378) | -2.15 (3.909)
  Frequency of itching due to AD Day 113: number analyzed (Participants) | 23 | 24 | 25 | 36 | 34
  Frequency of itching due to AD Day 113 | -2.00 (2.970) | -1.42 (3.035) | -1.04 (2.557) | -1.81 (3.188) | -1.50 (3.816)

12. Secondary Outcome: Percentage of Participants Achieving a >=50% Improvement in the EASI Total Score (EASI50) at All Scheduled Time Points
Description: as for outcome 5
Time Frame: All scheduled time points, including Weeks 1, 2, 4, 6, 8, 12, 13, 14, 16
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | PF-04965842 10mg QD | PF-04965842 30mg QD | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 56 | 49 | 51 | 56 | 55
percentage of participants
  Week 1: number analyzed (Participants) | 54 | 48 | 50 | 55 | 54
  Week 1 | 9.3 | 8.3 | 14.0 | 12.7 | 40.7
  Week 2: number analyzed (Participants) | 55 | 49 | 50 | 55 | 52
  Week 2 | 27.3 | 16.3 | 24.0 | 36.4 | 65.4
  Week 4: number analyzed (Participants) | 55 | 49 | 50 | 55 | 54
  Week 4 | 27.3 | 30.6 | 36.0 | 58.2 | 85.2
  Week 6: number analyzed (Participants) | 55 | 49 | 50 | 55 | 54
  Week 6 | 36.4 | 30.6 | 40.0 | 60.0 | 90.7
  Week 8: number analyzed (Participants) | 55 | 49 | 50 | 55 | 53
  Week 8 | 30.9 | 36.7 | 40.0 | 60.0 | 90.6
  Week 12: number analyzed (Participants) | 52 | 46 | 45 | 54 | 48
  Week 12 | 26.9 | 26.1 | 33.3 | 55.6 | 79.2
  Week 13: number analyzed (Participants) | 30 | 29 | 31 | 38 | 45
  Week 13 | 43.3 | 41.4 | 45.2 | 55.3 | 75.6
  Week 14: number analyzed (Participants) | 32 | 28 | 29 | 40 | 44
  Week 14 | 37.5 | 42.9 | 37.9 | 50.0 | 65.9
  Week 16: number analyzed (Participants) | 28 | 26 | 27 | 36 | 38
  Week 16 | 42.9 | 42.3 | 33.3 | 41.7 | 68.4

13. Secondary Outcome: Percentage of Participants Achieving a >=75% Improvement in the EASI Total Score (EASI75) at All Scheduled Time Points
Description: as for outcome 5
Time Frame: All scheduled time points, including Weeks 1, 2, 4, 6, 8, 12, 13, 14, 16
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | PF-04965842 10mg QD | PF-04965842 30mg QD | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 56 | 49 | 51 | 56 | 55
percentage of participants
  Week 1: number analyzed (Participants) | 54 | 48 | 50 | 55 | 54
  Week 1 | 3.7 | 2.1 | 6.0 | 3.6 | 16.7
  Week 2: number analyzed (Participants) | 55 | 49 | 50 | 55 | 52
  Week 2 | 5.5 | 12.2 | 6.0 | 12.7 | 36.5
  Week 4: number analyzed (Participants) | 55 | 49 | 50 | 55 | 54
  Week 4 | 10.9 | 18.4 | 20.0 | 27.3 | 57.4
  Week 6: number analyzed (Participants) | 55 | 49 | 50 | 55 | 54
  Week 6 | 16.4 | 18.4 | 18.0 | 38.2 | 68.5
  Week 8: number analyzed (Participants) | 55 | 49 | 50 | 55 | 53
  Week 8 | 20.0 | 22.4 | 22.0 | 40.0 | 73.6
  Week 12: number analyzed (Participants) | 52 | 46 | 45 | 54 | 48
  Week 12 | 15.4 | 17.4 | 13.3 | 40.7 | 64.6
  Week 13: number analyzed (Participants) | 30 | 29 | 31 | 38 | 45
  Week 13 | 26.7 | 27.6 | 12.9 | 36.8 | 55.6
  Week 14: number analyzed (Participants) | 32 | 28 | 29 | 40 | 44
  Week 14 | 31.3 | 25.0 | 6.9 | 35.0 | 45.5
  Week 16: number analyzed (Participants) | 28 | 26 | 27 | 36 | 38
  Week 16 | 32.1 | 38.5 | 3.7 | 25.0 | 36.8

14. Secondary Outcome: Percentage of Participants Achieving a >=90% Improvement in the EASI Total Score (EASI90) at All Scheduled Time Points
Description: as for outcome 5
Time Frame: All scheduled time points, including Weeks 1, 2, 4, 6, 8, 12, 13, 14, 16
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | PF-04965842 10mg QD | PF-04965842 30mg QD | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 56 | 49 | 51 | 56 | 55
percentage of participants
  Week 1: number analyzed (Participants) | 54 | 48 | 50 | 55 | 54
  Week 1 | 0.0 | 2.1 | 4.0 | 0.0 | 7.4
  Week 2: number analyzed (Participants) | 55 | 49 | 50 | 55 | 52
  Week 2 | 0.0 | 6.1 | 4.0 | 5.5 | 19.2
  Week 4: number analyzed (Participants) | 55 | 49 | 50 | 55 | 54
  Week 4 | 1.8 | 8.2 | 8.0 | 10.9 | 38.9
  Week 6: number analyzed (Participants) | 55 | 49 | 50 | 55 | 54
  Week 6 | 7.3 | 14.3 | 14.0 | 16.4 | 44.4
  Week 8: number analyzed (Participants) | 55 | 49 | 50 | 55 | 53
  Week 8 | 5.5 | 12.2 | 8.0 | 23.6 | 43.4
  Week 12: number analyzed (Participants) | 52 | 46 | 45 | 54 | 48
  Week 12 | 9.6 | 10.9 | 0.0 | 25.9 | 52.1
  Week 13: number analyzed (Participants) | 30 | 29 | 31 | 38 | 45
  Week 13 | 10.0 | 13.8 | 3.2 | 23.7 | 31.1
  Week 14: number analyzed (Participants) | 32 | 28 | 29 | 40 | 44
  Week 14 | 15.6 | 14.3 | 0.0 | 17.5 | 18.2
  Week 16: number analyzed (Participants) | 28 | 26 | 27 | 36 | 38
  Week 16 | 14.3 | 23.1 | 3.7 | 8.3 | 10.5

15. Secondary Outcome: Change From Baseline in Affected BSA at All Scheduled Time Points
Description: BSA Efficacy is derived from the sum of the BSA in handprints across 4 body regions assessed as part of the EASI assessment. Handprint refers to that of each individual participant for their own measurement. The BSA Efficacy ranges from 0 to 100%, with higher values representing greater severity of AD. Since the scalp, palms, and soles are excluded from the BSA (Efficacy) assessment, the maximum possible value is less than 100%.
Time Frame: Baseline and all scheduled time points, including Weeks 1, 2, 4, 6, 8, 12, 13, 14, 16
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of BSA
Arm/Group | Placebo | PF-04965842 10mg QD | PF-04965842 30mg QD | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 56 | 49 | 51 | 56 | 55
percentage of BSA
  Week 1: number analyzed (Participants) | 54 | 48 | 49 | 55 | 53
  Week 1 | -0.06 (6.699) | -3.76 (13.940) | -2.45 (7.017) | -4.63 (12.144) | -10.86 (15.690)
  Week 2: number analyzed (Participants) | 55 | 48 | 47 | 53 | 50
  Week 2 | -5.43 (10.030) | -4.84 (16.179) | -6.51 (10.485) | -10.80 (16.432) | -21.30 (19.285)
  Week 4: number analyzed (Participants) | 50 | 45 | 47 | 52 | 52
  Week 4 | -6.34 (16.138) | -8.93 (15.960) | -9.59 (14.845) | -17.77 (19.956) | -28.55 (20.447)
  Week 6: number analyzed (Participants) | 44 | 38 | 43 | 48 | 52
  Week 6 | -10.79 (16.413) | -11.80 (22.324) | -10.71 (15.007) | -18.80 (23.387) | -30.51 (20.853)
  Week 8: number analyzed (Participants) | 41 | 36 | 43 | 47 | 49
  Week 8 | -9.71 (17.837) | -12.98 (25.552) | -10.79 (19.259) | -19.41 (23.596) | -29.98 (20.864)
  Week 12: number analyzed (Participants) | 35 | 29 | 30 | 43 | 42
  Week 12 | -13.82 (22.348) | -11.59 (27.112) | -9.37 (18.783) | -22.21 (22.199) | -27.72 (18.361)
  Week 13: number analyzed (Participants) | 30 | 29 | 31 | 38 | 45
  Week 13 | -7.90 (18.233) | -11.07 (25.457) | -7.79 (17.469) | -17.88 (20.905) | -22.61 (22.390)
  Week 14: number analyzed (Participants) | 32 | 28 | 29 | 40 | 44
  Week 14 | -8.97 (16.223) | -10.46 (26.130) | -6.33 (17.404) | -12.75 (22.492) | -16.35 (18.931)
  Week 16: number analyzed (Participants) | 28 | 26 | 27 | 36 | 38
  Week 16 | -8.09 (15.797) | -14.64 (20.948) | -3.52 (20.967) | -5.55 (21.079) | -17.88 (17.059)

16. Secondary Outcome: Change From Baseline in Scoring Atopic Dermatitis (SCORAD) at All Scheduled Time Points
Description: SCORAD is a validated scoring index for AD, which combines extent (0-100), severity (0-18), and subjective symptoms (0-20) based on pruritus and sleep loss, each scored (0-10). Extent, denoted as A, is measured by BSA affected by AD as a percentage of the whole BSA. The score for each body region is added up to determine A (maximum of 100%). Severity, denoted as B, consists of the severity of several signs. Each is assessed as none(0), mild(1), moderate(2) or severe(3). The severity scores are added together to give B (maximum of 18). Subjective symptoms, denoted as C, are each scored by the subject or caregiver using a numeric rating scale (NRS) where "0" is no itch (or no sleeplessness) and "10" is the worst imaginable itch (or sleeplessness). These scores are added to give 'C' (maximum of 20). The SCORAD for an individual is calculated by the formula: A/5 + 7B/2 + C (can range from 0 to 103). Higher values of SCORAD represent worse outcome.
Time Frame: Baseline and all scheduled time points, including Weeks 1, 2, 4, 6, 8, 12, 13, 14, 16
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | PF-04965842 10mg QD | PF-04965842 30mg QD | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 56 | 49 | 51 | 56 | 55
units on a scale
  Week 1: number analyzed (Participants) | 54 | 48 | 49 | 55 | 53
  Week 1 | -7.910 (12.4625) | -5.000 (13.3310) | -8.388 (14.6316) | -12.024 (12.4053) | -21.326 (15.8867)
  Week 2: number analyzed (Participants) | 55 | 48 | 47 | 53 | 50
  Week 2 | -10.905 (15.4157) | -8.795 (16.3883) | -13.266 (14.5268) | -20.286 (15.2402) | -32.152 (14.4354)
  Week 4: number analyzed (Participants) | 50 | 45 | 47 | 52 | 52
  Week 4 | -14.555 (16.6414) | -14.116 (19.1643) | -15.496 (16.4795) | -28.058 (16.6775) | -39.567 (14.7328)
  Week 6: number analyzed (Participants) | 44 | 38 | 43 | 48 | 52
  Week 6 | -19.527 (16.7869) | -16.667 (21.8577) | -19.930 (17.5966) | -29.729 (21.6156) | -41.458 (14.3943)
  Week 8: number analyzed (Participants) | 41 | 36 | 43 | 47 | 49
  Week 8 | -19.052 (18.5735) | -18.853 (21.7947) | -19.534 (18.7098) | -30.148 (20.7887) | -42.604 (13.9771)
  Week 12: number analyzed (Participants) | 35 | 29 | 30 | 43 | 42
  Week 12 | -18.647 (20.0191) | -17.986 (23.1948) | -21.211 (17.6774) | -33.145 (21.4221) | -41.384 (15.4359)
  Week 13: number analyzed (Participants) | 30 | 29 | 31 | 38 | 45
  Week 13 | -16.603 (21.3850) | -16.895 (22.1132) | -15.023 (16.1573) | -24.261 (19.4912) | -29.884 (19.1501)
  Week 14: number analyzed (Participants) | 32 | 28 | 29 | 40 | 44
  Week 14 | -17.987 (22.0893) | -15.842 (19.5000) | -12.768 (13.6914) | -20.211 (20.2920) | -21.292 (17.7775)
  Week 16: number analyzed (Participants) | 28 | 26 | 27 | 36 | 38
  Week 16 | -19.408 (22.1744) | -18.925 (21.5459) | -12.716 (15.9390) | -17.753 (19.1842) | -21.024 (18.1576)

17. Secondary Outcome: Percent Change From Baseline in SCORAD at All Scheduled Time Points
Description: as for outcome 16
Time Frame: Baseline and all scheduled time points, including Weeks 1, 2, 4, 6, 8, 12, 13, 14, 16
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04965842 10mg QD | PF-04965842 30mg QD | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 56 | 49 | 51 | 56 | 55
percent change
  Week 1: number analyzed (Participants) | 54 | 48 | 49 | 55 | 53
  Week 1 | -11.547 (19.7128) | -7.287 (20.6403) | -13.068 (21.0746) | -19.185 (20.0094) | -34.660 (25.0837)
  Week 2: number analyzed (Participants) | 55 | 48 | 47 | 53 | 50
  Week 2 | -16.488 (23.0011) | -12.980 (25.5198) | -20.613 (21.0283) | -31.025 (23.9881) | -51.384 (21.3581)
  Week 4: number analyzed (Participants) | 50 | 45 | 47 | 52 | 52
  Week 4 | -22.476 (26.5163) | -20.751 (29.0846) | -24.866 (25.3755) | -43.846 (26.2001) | -63.970 (21.6701)
  Week 6: number analyzed (Participants) | 44 | 38 | 43 | 48 | 52
  Week 6 | -30.789 (27.9424) | -25.851 (34.2950) | -31.276 (29.6517) | -45.270 (34.3893) | -66.971 (22.4343)
  Week 8: number analyzed (Participants) | 41 | 36 | 43 | 47 | 49
  Week 8 | -29.624 (30.5625) | -28.599 (33.1460) | -30.480 (29.4742) | -46.187 (32.7984) | -69.736 (21.4403)
  Week 12: number analyzed (Participants) | 35 | 29 | 30 | 43 | 42
  Week 12 | -29.379 (31.9081) | -27.607 (36.5015) | -32.535 (25.2711) | -51.624 (33.0106) | -68.537 (24.2392)
  Week 13: number analyzed (Participants) | 30 | 29 | 31 | 38 | 45
  Week 13 | -26.794 (34.3384) | -26.905 (34.1879) | -24.232 (26.2461) | -38.193 (32.3458) | -48.428 (30.1133)
  Week 14: number analyzed (Participants) | 32 | 28 | 29 | 40 | 44
  Week 14 | -29.393 (36.6642) | -25.511 (31.1985) | -20.072 (21.7399) | -31.521 (34.1268) | -36.519 (28.5404)
  Week 16: number analyzed (Participants) | 28 | 26 | 27 | 36 | 38
  Week 16 | -31.972 (36.5058) | -30.135 (34.2361) | -19.794 (25.0550) | -29.130 (33.1868) | -34.995 (27.4996)

18. Secondary Outcome: Percentage of Participants Achieving a >=50% Improvement in SCORAD (SCORAD50) From Baseline at All Scheduled Time Points
Description: as for outcome 16
Time Frame: Baseline and all scheduled time points, including Weeks 1, 2, 4, 6, 8, 12, 13, 14, 16
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | PF-04965842 10mg QD | PF-04965842 30mg QD | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 56 | 49 | 51 | 56 | 55
percentage of participants
  Week 1: number analyzed (Participants) | 54 | 48 | 50 | 55 | 54
  Week 1 | 3.7 | 2.1 | 6.0 | 7.3 | 29.6
  Week 2: number analyzed (Participants) | 55 | 49 | 50 | 55 | 52
  Week 2 | 5.5 | 10.2 | 10.0 | 18.2 | 55.8
  Week 4: number analyzed (Participants) | 55 | 49 | 50 | 55 | 54
  Week 4 | 20.0 | 12.2 | 16.0 | 43.6 | 75.9
  Week 6: number analyzed (Participants) | 55 | 49 | 50 | 55 | 54
  Week 6 | 21.8 | 16.3 | 26.0 | 45.5 | 74.1
  Week 8: number analyzed (Participants) | 55 | 49 | 50 | 55 | 53
  Week 8 | 23.6 | 22.4 | 30.0 | 43.6 | 73.6
  Week 12: number analyzed (Participants) | 52 | 46 | 45 | 54 | 48
  Week 12 | 19.2 | 13.0 | 15.6 | 50.0 | 72.9
  Week 13: number analyzed (Participants) | 30 | 29 | 31 | 38 | 45
  Week 13 | 26.7 | 20.7 | 16.1 | 34.2 | 48.9
  Week 14: number analyzed (Participants) | 32 | 28 | 29 | 40 | 44
  Week 14 | 31.3 | 17.9 | 3.4 | 32.5 | 36.4
  Week 16: number analyzed (Participants) | 28 | 26 | 27 | 36 | 38
  Week 16 | 39.3 | 30.8 | 14.8 | 25.0 | 34.2

19. Secondary Outcome: Percentage of Participants Achieving a >=75% Improvement in SCORAD (SCORAD75) From Baseline at All Scheduled Time Points
Description: as for outcome 16
Time Frame: Baseline and all scheduled time points, including Weeks 1, 2, 4, 6, 8, 12, 13, 14, 16
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | PF-04965842 10mg QD | PF-04965842 30mg QD | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 56 | 49 | 51 | 56 | 55
percentage of participants
  Week 1: number analyzed (Participants) | 54 | 48 | 50 | 55 | 54
  Week 1 | 0.0 | 2.1 | 2.0 | 1.8 | 3.7
  Week 2: number analyzed (Participants) | 55 | 49 | 50 | 55 | 52
  Week 2 | 0.0 | 2.0 | 2.0 | 3.6 | 11.5
  Week 4: number analyzed (Participants) | 55 | 49 | 50 | 55 | 54
  Week 4 | 1.8 | 4.1 | 4.0 | 14.5 | 27.8
  Week 6: number analyzed (Participants) | 55 | 49 | 50 | 55 | 54
  Week 6 | 5.5 | 12.2 | 4.0 | 20.0 | 37.0
  Week 8: number analyzed (Participants) | 55 | 49 | 50 | 55 | 53
  Week 8 | 3.6 | 6.1 | 2.0 | 16.4 | 35.8
  Week 12: number analyzed (Participants) | 52 | 46 | 45 | 54 | 48
  Week 12 | 3.8 | 10.9 | 0.0 | 18.5 | 37.5
  Week 13: number analyzed (Participants) | 30 | 29 | 31 | 38 | 45
  Week 13 | 13.3 | 10.3 | 0.0 | 18.4 | 15.6
  Week 14: number analyzed (Participants) | 32 | 28 | 29 | 40 | 44
  Week 14 | 15.6 | 7.1 | 0.0 | 12.5 | 11.4
  Week 16: number analyzed (Participants) | 28 | 26 | 27 | 36 | 38
  Week 16 | 14.3 | 11.5 | 0.0 | 11.1 | 2.6

20. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a subject administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. Treatment-emergent AEs were events that occurred between the first dose of study drug and the subject's last visit (Week 16) that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline till Week 16
Population: Safety Analysis Set: All participants who received at least 1 dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-04965842 10mg QD | PF-04965842 30mg QD | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 56 | 49 | 51 | 56 | 55
participants | 32 | 34 | 34 | 43 | 41

21. Secondary Outcome: Number of Participants With Specific Clinical Laboratory Abnormalities (Anemia, Neutropenia, Thrombocytopenia, Lymphopenia, Lipid Profile, Liver Function Tests (LFTs)
Time Frame: Baseline up to Week 16
Population: Safety Analysis Set: All participants who received at least 1 dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-04965842 10mg QD | PF-04965842 30mg QD | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 56 | 49 | 51 | 56 | 55
participants
  AEs of anemia | 0 | 0 | 0 | 0 | 0
  AEs of neutropenia | 0 | 0 | 0 | 0 | 1
  AEs of thrombocytopenia | 0 | 0 | 0 | 0 | 1
  AEs of lymphopenia | 0 | 0 | 0 | 0 | 0
  AEs of lipid profile | 0 | 0 | 0 | 0 | 0
  AEs of liver function tests | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Percentage of Participants With Patient Global Assessment (PtGA) of AD of Clear (0) or Almost Clear (1) and >=2 Points Improvement From Baseline at All Scheduled Time Points
Description: The PtGA asked the participant to evaluate the overall cutaneous disease at that point in time on a single-item, 5-point scale. The same category labels used in the Physician's Global Assessment was used for the PtGA, ie, "severe (4)", "moderate (3)", "mild (2)","almost clear (1)", and "clear (0)". The PtGA was completed as per schedule of activities.
Time Frame: Baseline and all scheduled time points, including Weeks 1, 2, 4, 6, 8, 12, 14, 16
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | PF-04965842 10mg QD | PF-04965842 30mg QD | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 56 | 49 | 51 | 56 | 55
percentage of participants
  Week 1: number analyzed (Participants) | 53 | 48 | 49 | 53 | 54
  Week 1 | 0.0 | 2.1 | 4.1 | 1.9 | 16.7
  Week 2: number analyzed (Participants) | 54 | 49 | 49 | 54 | 52
  Week 2 | 5.6 | 0.0 | 6.1 | 16.7 | 32.7
  Week 4: number analyzed (Participants) | 53 | 49 | 49 | 54 | 53
  Week 4 | 3.8 | 6.1 | 8.2 | 22.2 | 54.7
  Week 6: number analyzed (Participants) | 53 | 49 | 49 | 54 | 54
  Week 6 | 3.8 | 10.2 | 8.2 | 22.2 | 51.9
  Week 8: number analyzed (Participants) | 54 | 49 | 49 | 54 | 53
  Week 8 | 1.9 | 6.1 | 6.1 | 24.1 | 56.6
  Week 12: number analyzed (Participants) | 54 | 48 | 48 | 54 | 52
  Week 12 | 7.4 | 12.5 | 0.0 | 25.9 | 51.9
  Week 14: number analyzed (Participants) | 31 | 29 | 28 | 38 | 45
  Week 14 | 3.2 | 10.3 | 0.0 | 15.8 | 15.6
  Week 16: number analyzed (Participants) | 27 | 26 | 26 | 34 | 38
  Week 16 | 11.1 | 7.7 | 0.0 | 11.8 | 10.5

23. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Total Score at All Scheduled Time Points
Description: The DLQI is a general dermatology questionnaire that consists of 10 items that assess participant health-related quality of life (daily activities, personal relationships, symptoms and feelings, leisure, work and school, and treatment). It has been extensively used in clinical trials for AD. The DLQI is a psychometrically valid and reliable instrument that has been translated into several languages, and the DLQI total scores have been shown to be responsive to change. The minimally important difference for the DLQI has been estimated as a 2-5 point change from baseline. Each item is scored as "very much (3)", "a lot (2)", "a little (1)" and "not at all (0)". The score can range from 0 to 30. The higher values represent the worse dermatology life quality.
Time Frame: Baseline and all scheduled time points, including Weeks 1, 2, 4, 6, 8, 12, 14, 16
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | PF-04965842 10mg QD | PF-04965842 30mg QD | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 56 | 49 | 51 | 56 | 55
units on a scale
  Week 1: number analyzed (Participants) | 53 | 48 | 48 | 54 | 53
  Week 1 | -1.4 (6.04) | -1.4 (5.66) | -3.4 (6.28) | -5.1 (5.40) | -6.3 (5.55)
  Week 2: number analyzed (Participants) | 53 | 48 | 46 | 52 | 50
  Week 2 | -2.3 (5.42) | -1.9 (6.58) | -5.0 (5.55) | -7.5 (6.39) | -8.6 (6.46)
  Week 4: number analyzed (Participants) | 48 | 45 | 45 | 51 | 51
  Week 4 | -2.6 (6.77) | -3.7 (7.33) | -4.7 (5.62) | -8.2 (7.48) | -9.7 (6.82)
  Week 6: number analyzed (Participants) | 42 | 38 | 42 | 47 | 52
  Week 6 | -4.2 (6.01) | -4.6 (7.30) | -4.1 (7.75) | -9.1 (6.75) | -10.2 (6.72)
  Week 8: number analyzed (Participants) | 40 | 36 | 42 | 46 | 49
  Week 8 | -3.7 (7.67) | -5.6 (8.44) | -4.8 (8.52) | -9.2 (7.95) | -9.8 (7.10)
  Week 12: number analyzed (Participants) | 36 | 31 | 33 | 43 | 46
  Week 12 | -4.6 (8.49) | -4.5 (8.90) | -5.2 (7.30) | -9.8 (8.18) | -9.5 (7.28)
  Week 14: number analyzed (Participants) | 31 | 29 | 28 | 39 | 45
  Week 14 | -3.1 (8.24) | -3.9 (7.62) | -3.6 (6.60) | -6.2 (7.87) | -4.4 (8.78)
  Week 16: number analyzed (Participants) | 27 | 26 | 26 | 34 | 38
  Week 16 | -4.5 (7.95) | -4.5 (7.14) | -3.5 (7.17) | -4.6 (7.62) | -3.6 (7.39)

24. Secondary Outcome: Change From Baseline in Patient Oriented Eczema Measure (POEM) at All Scheduled Time Points
Description: The POEM is a 7-item patient reported outcome (PRO) measure used to assess the impact of AD over the past week. Each item is scored as "no days (0)", "1-2 days (1)", "3-4 days (2)", "5-6 days (3)" and "every day (4)". The score ranges from 0 to 28. The higher values represent more severe AD.
Time Frame: Baseline and all scheduled time points, including Weeks 1, 2, 4, 6, 8, 12, 14, 16
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | PF-04965842 10mg QD | PF-04965842 30mg QD | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 56 | 49 | 51 | 56 | 55
units on a scale
  Week 1: number analyzed (Participants) | 53 | 48 | 48 | 53 | 50
  Week 1 | -1.1 (3.59) | -0.6 (4.17) | -2.1 (5.83) | -3.9 (4.67) | -9.2 (5.77)
  Week 2: number analyzed (Participants) | 51 | 48 | 45 | 50 | 50
  Week 2 | -2.2 (4.20) | -1.9 (6.13) | -4.1 (6.04) | -7.2 (6.79) | -11.9 (5.95)
  Week 4: number analyzed (Participants) | 48 | 45 | 44 | 50 | 50
  Week 4 | -2.2 (6.05) | -3.6 (6.35) | -4.3 (5.69) | -8.7 (8.30) | -14.6 (6.20)
  Week 6: number analyzed (Participants) | 41 | 38 | 42 | 45 | 50
  Week 6 | -3.5 (5.24) | -4.3 (7.63) | -3.9 (7.43) | -10.4 (8.17) | -15.0 (5.92)
  Week 8: number analyzed (Participants) | 40 | 36 | 42 | 45 | 48
  Week 8 | -2.3 (5.91) | -4.3 (8.94) | -5.4 (8.05) | -10.6 (8.47) | -15.2 (6.15)
  Week 12: number analyzed (Participants) | 36 | 31 | 33 | 41 | 45
  Week 12 | -3.8 (8.21) | -4.7 (8.83) | -5.3 (7.60) | -11.4 (8.08) | -15.1 (6.99)
  Week 14: number analyzed (Participants) | 31 | 29 | 28 | 38 | 44
  Week 14 | -2.2 (6.45) | -3.9 (8.04) | -2.7 (6.05) | -6.3 (7.12) | -6.2 (6.97)
  Week 16: number analyzed (Participants) | 27 | 26 | 26 | 34 | 37
  Week 16 | -3.0 (7.76) | -3.0 (7.67) | -2.2 (6.80) | -4.3 (6.20) | -5.9 (5.93)

25. Secondary Outcome: Change From Baseline in the Hospital and Anxiety Depression Scale (HADS) at All Scheduled Time Points
Description: The HADS is a 14-item PRO measure used to detect states of anxiety and depression over the past week. The HADS was completed as per schedule of activities. Seven of the items relate to anxiety and seven relate to depression. Each item is scored from 0 to 3 which means a person can score between 0 to 21 for either anxiety or depression. Higher values represent worse outcome.
Time Frame: Baseline and all scheduled time points, including Weeks 1, 2, 4, 6, 8, 12, 14, 16
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | PF-04965842 10mg QD | PF-04965842 30mg QD | PF-04965842 100mg QD | PF-04965842 200mg QD
Number analyzed (Participants) | 56 | 49 | 51 | 56 | 55
units on a scale
  Depression score Week 1: number analyzed (Participants) | 53 | 48 | 48 | 54 | 53
  Depression score Week 1 | -0.5 (2.71) | 0.0 (2.38) | -0.6 (2.49) | -0.9 (2.94) | -1.0 (2.16)
  Depression score Week 2: number analyzed (Participants) | 53 | 48 | 46 | 52 | 50
  Depression score Week 2 | -0.5 (2.78) | 0.4 (2.99) | -1.1 (1.85) | -1.2 (2.93) | -1.8 (2.66)
  Depression score Week 4: number analyzed (Participants) | 47 | 45 | 45 | 51 | 51
  Depression score Week 4 | -0.5 (3.00) | -0.4 (3.26) | -0.8 (2.05) | -1.5 (3.35) | -2.1 (3.30)
  Depression score Week 8: number analyzed (Participants) | 41 | 36 | 42 | 46 | 50
  Depression score Week 8 | -0.7 (3.31) | -1.3 (3.76) | -0.9 (2.84) | -2.1 (3.35) | -1.7 (3.08)
  Depression score Week 12: number analyzed (Participants) | 36 | 31 | 33 | 43 | 46
  Depression score Week 12 | -0.9 (3.96) | -0.9 (3.65) | -0.5 (2.83) | -2.4 (3.74) | -1.8 (3.90)
  Depression score Week 14: number analyzed (Participants) | 31 | 29 | 28 | 39 | 45
  Depression score Week 14 | 0.1 (3.41) | -1.2 (3.50) | -0.9 (1.53) | -1.7 (4.31) | -0.1 (4.18)
  Depression score Week 16: number analyzed (Participants) | 27 | 26 | 26 | 34 | 38
  Depression score Week 16 | -0.7 (3.18) | -1.1 (3.59) | -1.0 (1.85) | -1.4 (3.93) | -0.1 (3.57)
  Anxiety score Week 1: number analyzed (Participants) | 53 | 48 | 48 | 54 | 53
  Anxiety score Week 1 | -1.0 (2.66) | 0.2 (2.41) | -0.2 (2.49) | -1.1 (2.26) | -1.2 (2.71)
  Anxiety score Week 2: number analyzed (Participants) | 53 | 48 | 46 | 52 | 50
  Anxiety score Week 2 | -1.5 (2.87) | -0.4 (2.56) | -0.9 (2.88) | -1.7 (2.81) | -2.4 (3.15)
  Anxiety score Week 4: number analyzed (Participants) | 47 | 46 | 45 | 51 | 51
  Anxiety score Week 4 | -1.6 (3.18) | -1.0 (2.80) | -0.7 (2.69) | -1.7 (2.95) | -2.4 (4.04)
  Anxiety score Week 8: number analyzed (Participants) | 41 | 36 | 42 | 46 | 50
  Anxiety score Week 8 | -1.7 (2.33) | -1.6 (2.67) | -1.4 (3.21) | -2.7 (3.44) | -2.5 (3.31)
  Anxiety score Week 12: number analyzed (Participants) | 36 | 31 | 33 | 43 | 46
  Anxiety score Week 12 | -2.6 (3.01) | -1.5 (2.85) | -1.0 (3.43) | -2.8 (3.71) | -2.5 (3.51)
  Anxiety score Week 14: number analyzed (Participants) | 31 | 29 | 28 | 39 | 45
  Anxiety score Week 14 | -2.3 (3.43) | -1.5 (3.17) | -1.4 (2.96) | -2.0 (3.49) | -1.5 (3.93)
  Anxiety score Week 16: number analyzed (Participants) | 27 | 26 | 26 | 34 | 38
  Anxiety score Week 16 | -2.9 (3.75) | -2.2 (3.38) | -0.7 (3.27) | -1.4 (3.85) | -1.5 (3.10)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 16
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Placebo | PF-04965842 10mg QD | PF-04965842 30mg QD | PF-04965842 100mg QD | PF-04965842 200mg QD
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/49 | 0/51 | 0/56 | 0/55
Serious Adverse Events (participants affected / at risk) | 2/56 | 2/49 | 0/51 | 3/56 | 2/55
Other Adverse Events (participants affected / at risk) | 17/56 | 18/49 | 25/51 | 25/56 | 27/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=56) | PF-04965842 10mg QD (N=49) | PF-04965842 30mg QD (N=51) | PF-04965842 100mg QD (N=56) | PF-04965842 200mg QD (N=55)
Eczema herpeticum (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=56) | PF-04965842 10mg QD (N=49) | PF-04965842 30mg QD (N=51) | PF-04965842 100mg QD (N=56) | PF-04965842 200mg QD (N=55)
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 1 | 1 | 5
Nausea (Gastrointestinal disorders) | 1 | 3 | 3 | 1 | 8
Upper respiratory tract infection (Infections and infestations) | 5 | 3 | 5 | 3 | 5
Viral upper respiratory tract infection (Infections and infestations) | 5 | 5 | 6 | 10 | 7
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 3
Headache (Nervous system disorders) | 2 | 2 | 5 | 5 | 4
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 6 | 8 | 9 | 7 | 7
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-05-09): https://cdn.clinicaltrials.gov/large-docs/67/NCT02780167/SAP_000.pdf
  • Study Protocol (2015-12-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT02780167/Prot_001.pdf